

Paritaprevir/r – ombitasvir and dasabuvir P16-014 Protocol

# **Title Page**

| Title | Real World Evidence of the Effectiveness of Paritaprevir/r – Ombitasvir, ± Dasabuvir, ± Ribavirin and Patient Support Program in Patients with <b>C</b> hronic Hepatitis C - An Obse <b>r</b> vat <b>ion</b> al Study in Isra <b>e</b> l (CITRINE STUDY) |
|---|---|
| Protocol Version Identifier | Protocol Version 1, 16 Mar 2016 |
| Date of Last Version of Protocol | Not Applicable |
| Research Question and Objectives | What is the effectiveness of the interferon-free regimen of Paritaprevir/r – Ombitasvir, ± Dasabuvir, ± Ribavirin and Patient Support Program and its influence on patients with CHC in a real life setting across clinical practice patient populations? |
| Country(-ies) of Study | Israel |
| Main Author | |
| Marketing Authorization Holder(s) | AbbVie Ltd. |

This study will be conducted in compliance with this protocol and all applicable local regulatory requirements

| 1.0 | Table of Contents | |
|--------------------|----------------------------------|----|
| 1.0 | Table of Contents | 2 |
| 2.0 | Abbreviations | 5 |
| 3.0 | Responsible Parties | 8 |
| 4.0 | Abstract | |
| 5.0 | Amendments and Updates | 13 |
| 6.0 | Milestones | |
| 7.0 | Rationale and Background | 13 |
| 7.1 | Background | |
| 7.2 | Rationale | 19 |
| 8.0 | Research Question and Objectives | 20 |
| 8.1 | Research Question | 20 |
| 8.2 | Objectives | 20 |
| 8.2.1 | Primary Objective | 20 |
| 8.2.2 | Secondary Objectives | 21 |
| 9.0 | Research Methods | 21 |
| 9.1 | Study Design | 21 |
| 9.2 | Setting | 22 |
| 9.2.1 | Target Population | 22 |
| 9.2.2 | Study Duration | 23 |
| 9.2.3 | Termination Criteria | 23 |
| 9.2.4 | Investigator Selection Criteria | 23 |
| 9.3 | Variables | 24 |
| 9.3.1 | Primary Variable | 24 |
| 9.3.2 | Secondary Variables | 24 |
| 9.4 | Data Sources | 24 |
| 9.4.1 | Data to be Documented | 24 |
| 9.4.1.1 | Inclusion Documentation | 25 |
| | inclusion Documentation | |
| 9.4.1.2 | During Treatment Documentation | 26 |
| 9.4.1.2<br>9.4.1.3 | | |
| | During Treatment Documentation | 27 |

| 9.4.1.6 | Standardized Assessment Tools | |
|---|---|---|
| 9.5 | Study Size | |
| 9.6 | Data Management | 30 |
| 9.6.1 | Electronic Case Report Forms | 30 |
| 9.6.2 | Assignment of Preferred Terms | |
| 9.7 | Data Analysis | 32 |
| 9.7.1 | Analysis Population, Time Windows and Handling of Missing Data | 32 |
| 9.7.2 | Demographics and Disease Characteristics | |
| 9.7.3 | Effectiveness Analysis | |
| 9.7.3.1 | Primary Effectiveness Endpoint | |
| 9.7.3.2 | Secondary Effectiveness Endpoints | |
| 9.7.3.3 | Statistical Methods for Analysis of Effectiveness Variables | |
| 9.7.4 | Clinical Laboratory Data | |
| 9.7.5 | PSP and PAM | |
| 9.7.6 | Tolerability Analysis | 37 |
| 9.7.7 | Interim Assessments | |
| 9.8 | Quality Control | 38 |
| 9.9 | Limitations of the Research Methods | 38 |
| 10.0 | Protection of Human Subjects | 39 |
| 11.0 | Management and Reporting of Complaints | 39 |
| 11.1 | Medical Complaints | |
| 11.1.1 | Adverse Event Definition and Serious Adverse Event Categories | 40 |
| 11.1.2 | Severity | 42 |
| 11.1.3 | Relationship to Pharmaceutical Product | 42 |
| 11.1.4 | Serious Adverse Event Collection Period | 42 |
| 11.1.5 | Serious and non-serious Adverse Event Reporting | 43 |
| 11.1.6 | Pregnancy Reporting | 43 |
| 11.2 | Product Complaint | 43 |
| 11.2.1 | Definition | 43 |
| 11.2.2 | Reporting | 44 |
| 12.0 | Plans for Disseminating and Communicating Study Results | |

| 13.0 | References | |
|---|---|---|
| Annex 1. | Contact Insignia Health at www.insigniahealth.com | |
| | | DRAFT Version 0:03/08A t |
| | •••••• | 51 |
| Annex 2. | Patient Support Program (PSP) Utilization | |
| | Questionnaire | 52 |
| Annex 3. | Patient Support Program (PSP) Utilization and Sa- | |
| | tisfaction Questionnaire | 53 |
| Annex 4. | Child-Pugh Classification of Severity of Cirrhosis | 55 |
| 14.0 | Protocol Signature Page | 56 |

### 2.0 Abbreviations

AE adverse event

APRI AST to platelet ratio index

AFP alfa fetoprotein

ALT alanine-aminotransferase
AST aspartate-aminotransferase

ABBVIE Paritaprevir/r – ombitasvir ± dasabuvir

**REGIMEN** 

ANCOVA analysis of covariance

BMI body mass index
CA competent authority

CD4 cluster of differentiation 4

CHC chronic hepatitis C
CI confidence interval

CNI calcineurin

CP core population

CPFSU core population with sufficient follow-up data

CT computer tomography

DAA direct-acting antiviral agent

DDI drug-drug interaction

EC ethics committee

EDC electronic data capture

eCRF electronic case report form

EMA European Medicines Agency

EoT end of treatment

FDA Food and Drug Administration

FIB-4 Fibrosis-4 Score/Index

γ-GT gamma-glutamyltransferase

HCC hepatocellular carcinoma

HCP health care provider

Hb hemoglobin

HbA1c hemoglobin A1c
HBV hepatitis B virus
HCV hepatitis C virus

HDL high-density lipoprotein

HIV human immunodeficiency virus
HOMA homeostasis model assessment
HVPG hepatic venous pressure gradient

ICMJE International Committee of Medical Journal Editors

IEC/IRB independent ethics committee/- review board

IgA Immunoglobulin A
IgG Immunoglobulin G
IgM Immunoglobulin M

INN international non-proprietary name

INR international normalized ratio

LDL low-density lipoprotein LLoD lower limit of detection

LLoQ lower limit of quantification

MAH Marketing Authorization Holder

MedDRA Medical Dictionary for Regulatory Activities

MLR multiple logistic regression
MRI magnetic resonance imaging

NCP non-core population

NS3/NS4A nonstructural protein 3/nonstructural protein 4A

NS5A nonstructural protein 5A NS5B nonstructural protein 5B

OATP organic anion-transporting polypeptide

OLT orthotopic liver transplant

PAM-13 Patient Activation Measure 13

PCR polymerase chain reaction

pegIFN pegylated interferon

PRO patient reported outcome
PSP patient support program

PT preferred term

RBV ribavirin

RF rheumatoid factor
RNA ribonucleic acid

SAE serious adverse event SAP statistical analysis plan

SD standard deviation

SDP study designated physician

SNP single nucleotide polymorphism

SOC system organ class
SP safety population

SVR sustained virological response
SVR12 SVR at 12 weeks after EoT
SVR24 SVR at 24 weeks after EoT

TAI total activity impairment

TP target population

TWP total work productivity impairment

VAS visual analogue scale

WHO World Health Organization

# 3.0 Responsible Parties

Study Designated Physician (SDP):



### **Protocol Authors:**



### Vendor:

IST GmbH, Soldnerstrasse 1, D-68219 Mannheim, Germany www.istgmbh.com

### 4.0 Abstract

#### Title:

Real World Evidence of the Effectiveness of Paritaprevir/r – Ombitasvir, ± Dasabuvir, ± Ribavirin and Patient Support Program in Patients with Chronic Hepatitis C An Observational Study in Israel (CITRINE STUDY)

#### Rationale and Background:

The interferon-free combination regimen of Paritaprevir/r – ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) for the treatment of chronic hepatitis C (CHC) has been shown to be safe and effective in randomized controlled clinical trials with strict inclusion and exclusion criteria under well controlled conditions.

The ABBVIE REGIMEN is available in Israel for the treatment of CHC since 2015.

The rationale for this observational study is to determine how the efficacy and safety of the ABBVIE REGIMEN as demonstrated in pivotal trials translates into real world everyday clinical settings, which means evaluating its effectiveness. Whereas efficacy can be defined as a measure of the capacity of a treatment to produce the desired effect in a controlled environment, such as in a randomized controlled trial, effectiveness is the extent to which a drug achieves its intended effect in the usual clinical setting. Effectiveness trials typically have limited exclusion criteria and will involve the broader patient populations in routine clinical practice and per local label which might include patients with heterogenous compliance patterns and patients with significant comorbid conditions and could be used to model and disseminate best practices. Effectiveness research allows for external patient-, provider-, and system-level factors and can therefore be more relevant for health-care decisions by both providers in practice and policy-makers.

This observational study is the first effectiveness research examining the ABBVIE REGIMEN ± RBV, used according to local label, under real world conditions in Israel in a clinical practice patient population.

During the last decade when dual therapy with pegylated interferon (pegIFN) plus RBV was standard of care for the treatment of CHC, the discovery of predictive factors for virological response and the subsequent development of treatment algorithms marked a milestone in patient care for CHC. As a consequence, treatment could be effectively targeted to patients most likely to respond. Interestingly, many of the now well established predictors of response to pegIFN/RBV and first generation direct acting anitvirals (DAAs) in combination with pegIFN/RBV were not predictive of outcome in the development trials of the ABBVIE REGIMEN  $\pm$  RBV. This observational study may play an important part in bridging the data gaps. It may help identify predictive factors of response that are important in real world treatment settings and thus, could assist in further optimizing treatment with the interferon-free ABBVIE REGIMEN  $\pm$  RBV in the future.

The label of the ABBVIE REGIMEN ± RBV will vary according to hepatitis C virus (HCV) genotype/subtype and stage of liver disease. It is therefore relevant to understand the pattern of use and outcome in daily clinical practice. In addition, this study will provide data on the impact

of adherence on treatment outcomes in everyday settings, which may help treating physicians to improve the management of patients under their care.

The aim of this observational study is to provide evidence of the effectiveness of the interferonfree regimen of Paritaprevir/r – Ombitasvir, ± Dasabuvir, ± Ribavirin and PSP and its influence on patients with CHC in a real world setting across clinical practice patient populations.

#### **Research Question and Objectives:**

What is the effectiveness of the interferon-free regimen of Paritaprevir/r – Ombitasvir, ± Dasabuvir, ± Ribavirin and Patient Support Program and its influence on patients with CHC in a real life setting across clinical practice patient populations?

#### Primary Objective

 To describe in routine clinical practice the effectiveness of the interferon-free ABBVIE REGIMEN ± RBV in patients with CHC as evidenced by sustained virological response at 12 weeks after end of treatment (SVR12)

#### Secondary Objectives

- 2. To provide real world evidence for predictive factors of virological response
- 3. To describe the pattern of real world use of the ABBVIE REGIMEN  $\pm$  RBV with respect to different patient and treatment characteristics
- 4. To evaluate the contribution of the patient support program (PSP) to disease control, treatment continuation over time, patient satisfaction and PSP utilization
- 5. To describe the effect of the ABBVIE REGIMEN ± RBV on metabolic profile
- 6. To evaluate the effect of the ABBVIE REGIMEN ± RBV on extrahepatic manifestations and associated diseases like cryoglobulinemia/cutaneous vasculitis or porphyria cutanea tarda

#### Study Design:

This is a prospective, multi-center observational study in patients receiving the interferon-free ABBVIE REGIMEN ± RBV.

The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice and label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.

### **Target Population:**

Patients are eligible for observation in this cohort if the following applies:

- Treatment-naïve or -experienced adult male or female patients with confirmed CHC, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV according to standard of care and in line with the current local label
- If RBV is co-administered with the ABBVIE REGIMEN, it has been prescribed in line
  with the current local label (with special attention to contraception requirements and
  contraindication during pregnancy)
- Patients must voluntarily sign and date an informed consent form to use and/or disclose his/her anonymized health data prior to inclusion into the study
- Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial

#### Variables:

#### Primary Variable

The percentage of patients achieving SVR12 (HCV RNA <50 IU/mL 12 weeks [i.e. ≥70] days] after the last actual dose of the ABBVIE REGIMEN)

### Secondary Variables

- Type of treatment regimen (± Dasabuvir, ± RBV, intended and actual combination, dose and duration)
- PAM-13, PSP satisfaction and utilization questionnaires
- Metabolic laboratory profile (see section 9.4.1.1) prior to treatment initiation, and at all subsequent visits
- Cryoglobulins, immunoglobulins and porphyrin prior to treatment initiation, and at all subsequent visits

#### **Data Sources:**

Source documents are defined as original documents. The investigator will document patient data in his/her own patient files which will serve as source data for the study.

#### Study Size:

In phase III studies investigating the interferon-free ABBVIE REGIMEN ± RBV, SVR12 rates of at least 90% were observed, even in difficult-to-treat CHC patients (e.g. cirrhotic G1a treatment experienced patients). To describe in routine clinical practice the effectiveness of the ABBVIE REGIMEN ± RBV in patients with CHC, a precise estimate of the SVR12 rates should be achieved.

It is expected, that during the planned inclusion period of 8 months about 250 patients treated with the ABBVIE REGIMEN ± RBV can be included. It is furthermore, expected, that the number of patients to exclude from the core population will be not higher than 5-10%. With 235 evaluable patients the width of the 95% confidence interval (CI) will be 7.7% and 5.7% for SVR12 rates of 90% and 95%, respectively. If only 200 patients can be evaluated, the 95% CI will have a width of less than 8.4% for a SVR12 rate of at least 90% and less than 6.2% for a SVR12 rate of at least 95%.

#### Data Analysis:

The core population (CP) is defined as all patients of the target population (TP) (definition see above), who have started the treatment combination recommended in the current local label for their disease characteristics. Patients not receiving the treatment recommended in the local label will be summarized in the non-core population (NCP). In addition, the core population with sufficient follow-up data (CPSFU) is defined as all CP patients, who have (i) evaluable HCV RNA data ≥70 days after the last actual dose of the ABBVIE REGIMEN or (ii) a HCV RNA value ≥50 IU/mL at the last measurement or (iii) had HCV RNA <50 IU/mL at the last measurement, but no HCV RNA measurement ≥70 days after the last actual dose of the ABBVIE REGIMEN due to reasons related to safety (e.g. dropped out due to adverse event) or incomplete efficacy information (e.g. virologic failure such as relapse is reported in the electronic case report form (eCRF) but date and value of the corresponding HCV RNA test is missing). The safety population (SP) is defined as all patients who received at least one dose of the ABBVIE REGIMEN.

Descriptive and exploratory statistical methods will be used to analyze the data of the study. All baseline and disease characteristics will be summarized for the CP stratified by the CP analysis groups (based on genotype and fibrosis status), which are relevant for the scheduled treatment

combination. In addition, baseline summaries will be repeated for the SP and TP. Further details of analysis populations and the CP analysis groups will be specified in the statistical analysis plan (SAP).

The primary effectiveness analysis will be performed for CP patients, stratified by the CP analysis groups. Response rates (i.e. SVR12 rate, end of treatment [EoT] response rate, relapse rate, viral breakthrough) will be determined for the various CP analysis groups. The relapse rates will be estimated in patients of the CP analysis groups with EoT response and sufficient HCV RNA measurements post treatment. Viral breakthrough rates will be estimated in all patients of the CP analysis groups, who have at least one undetectable HCV RNA measurement on treatment and at least one on-treatment or EoT measurement thereafter. For all rates specified above 95%-confidence intervals (CIs) will be determined using the Wilson Score method.

Univariate and multiple logistic regression (MLR) methods will be used to investigate the impact of various explanatory covariates (e.g. demographic and disease characteristics, co-morbidities, type of treating institution, and prior treatment for CHC and response outcome in treatment experienced patients) on SVR12. These analyses will be of exploratory nature, data driven, and could be performed for various CP analysis groups since not each covariate might be predictive in each patient group. Furthermore, the fact that treatment regimens will differ in the various patient groups has to be taken into account, when selecting the patient groups for each MLR analysis. Backward selection procedures will be applied to generate the final MLR models and a p-value <0.05 will be used for the covariates to stay in the model in a backward elimination step. Logistic regression methods will also be used to investigate the impact of treatment adherence on SVR12.

All safety variables will be summarized for patients in the SP using descriptive statistical methods stratified by the type of combination treatment.

Milestones:

Start of Data Collection:

End of Data Collection:

Jun 2016

Jan 2018

Final Report of Study Results:

Dec 2018

### 5.0 Amendments and Updates

None

### 6.0 Milestones

Start of Data Collection: June 2016
 End of Data Collection: Jan 2018
 Final Report of Study Results: Dec 2018

### 7.0 Rationale and Background

### 7.1 Background

Infection with the hepatitis C virus (HCV) is associated with considerable morbidity and mortality [1] and is a leading cause of chronic liver disease, cirrhosis, and hepatocellular carcinoma (HCC), as well as the most common indication for liver transplantation in many countries [2]. Around 60-85% of subjects exposed to HCV do not clear the virus and go on to develop chronic disease [3] [4]. Chronic hepatitis C (CHC) affects an estimated 2-3% of the world's population - equaling approximately 130-210 million individuals [5] [6]. The prevalence varies markedly from one geographic area to another ranging from 0.1-1% in Western Europe to 1-2% in Latin America and up to 4.9% in some regions of Eastern Europe [7] [8] [9] [10].

HCV demonstrates a high degree of genetic variability and has been classified into seven major genotypes (and a large number of subtypes) the distribution of which varies globally [11]. Genotypes 1 through 3 are found worldwide; the other genotypes have a more restricted distribution, genotype 4 is found predominantly in the Middle East, Central Africa, and Egypt; genotype 5 in South Africa; and genotype 6 mainly in Asia. HCV genotypes 1a and 1b are the most common forms, accounting for 60% of HCV infections worldwide [12] [13] [14] [15].

HCV is primarily transmitted by parenteral exposures to contaminated blood, most frequently by injection drug use, exposures in health-care settings and inadequate infection-control practices (tattoo, piercing). Occupational, perinatal and sexual exposure can also result in transmission of HCV [16] [17]. Since the early 1990's routine blood screening protocols have been introduced in most countries and as a consequence

transmission of the virus is rarely seen following receipt of blood, blood products or through organ transplants.

The natural course of CHC leads to progressive fibrosis and can eventually lead to cirrhosis of the liver over the course of 20-30 years in approximately 15-30% of infected individuals [18]. Once patients become cirrhotic, around 6% per year are expected to develop hepatic decompensation (ascites, encephalopathy, variceal hemorrhage, hepatorenal syndrome, or hepatic synthetic dysfunction) and around 3% per year will develop HCC [19]. Over the same time frame, between 4 and 5% of patients can be expected to require liver transplantation or die [19] [20]. Progression is not necessarily a linear process and can be accelerated by a number of factors including the age of the patient, duration of HCV infection, male gender, alcohol consumption and co-infection with other viruses such as hepatitis B virus (HBV) and human immunodeficiency virus (HIV) [4] but also by concomitant steatosis and obesity. Comorbid conditions can impact CHC treatment eligibility, safety, tolerability and efficacy of therapy [21] [22].

The burden of advanced liver disease varies widely across countries and is dependent upon several factors including chronic HCV prevalence and age distribution (and duration of infection) of those infected [23]. Due to an aging cohort of patients and an associated increase in the incidence of severe liver disease, the burden of CHC will continue to increase. In persons 30–49 years of age, the prevalence of the disease is 3–fold higher than in other age groups. By 2020, the rates of HCC and liver-related deaths among individuals with CHC are expected to increase by 81% and 180%, respectively [24].

The eradication of the virus, defined as the absence of HCV ribonucleic acid (RNA) in serum (as shown by a sensitive test) at the end of treatment (EoT) and 12-24 weeks later (sustained virological response [SVR]), is the therapeutic goal of CHC treatment [25] [26] [27] and is generally accepted as a virological cure, thus, eventually preventing the aforementioned complications [26] [27].

Achieving an SVR was associated with significant reduction in all-cause death compared to patients who did not achieve SVR (5-year mortality rate in HCV genotype 1-infected patients: 6.7% vs 14.4%, respectively) [28]. In another study the 10-year cumulative all-cause mortality rate was 8.9% in patients with SVR and 26.0% without SVR (p<0.001), the liver-related mortality or transplantation was 1.9% with SVR and 27.4% without SVR (p<0.001), the rate of HCC was 5.1% with and 21.8% without SVR (p<0.001), and the rate of patients experiencing liver failure was 2.1% with and 29.9% (p<0.001) without SVR [29]. Patients with SVR following treatment with pegylated interferon (pegIFN) with or without RBV have also shown improvement in liver histology and a reduction in liver-related death in several studies [30] [31] [32]. Moreover, patients with compensated

cirrhosis who achieve SVR essentially eliminate their subsequent risk of decompensation, may achieve histologic regression, and decrease their risk of HCC by two-thirds [33] [34] [35].

In the 1980's and 1990's interferon alfa was the first drug to show activity against HCV. However, the effectiveness of interferon monotherapy in the treatment of CHC infection was generally unsatisfactory resulting in an overall SVR rate across genotypes of <20% [36] [37]. Combination therapy with interferon plus ribavirin (RBV) improved SVR rates but still overall rates across genotypes remained below 50% [38] [39]. Following the introduction of long-acting interferons (peginterferon alfa-2a and peginterferon alfa-2b [i.e. pegIFNs]) in combination with RBV more than a decade ago, further advances have been made in efficacy with overall rates of SVR up to 54-63% [39] [40] [41]. SVR rates vary substantially by HCV genotype with genotype 1 being the most difficult-to-treat, thus requiring longer treatment periods to obtain SVR with interferon-based dual therapy. SVR rates up to around 50% can be achieved in patients with genotype 1 whereas for genotypes 2 and 3 cure rates of up to 80% can be achieved [41].

Treatment with pegIFN and RBV is associated with considerable, often treatment-limiting toxicities including cytopenias, neuro-psychiatric disorders and influenza-like symptoms.

In 2011 the first direct-acting antivirals (DAAs), specifically the protease inhibitors boceprevir and telaprevir, have been approved by the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA) for treatment of HCV genotype 1. These first generation DAAs have significantly improved efficacy with rates of SVR reported as high as 63-75% among treatment-naïve HCV genotype 1 individuals [42] [43] [44]. However, these DAAs must be used in combination with pegIFN and RBV as triple combination therapy and the tolerability profile is further impaired by additional DAA specific adverse effects such as rash, pruritus, dysgeusia and anemia [42] [43] [44]. Treatment regimens with these DAAs are rather complicated with the necessity of futility rules and a response guided therapy duration of up to 48 weeks in selected patients.

Since 2014 the new standard of care for genotype 1 is pegIFN and RBV combined with either the nonstructural protein 3/nonstructural protein 4A (NS3/4A) protease inhibitor simeprevir or the nucleotide nonstructural protein 5B (NS5B) polymerase inhibitor sofosbuvir [45] [46].

Simeprevir is a NS3/4A protease inhibitor which was approved by the FDA at the end of 2013 and by the EMA in May 2014. In the phase III studies QUEST 1 and 2 treatment-naïve patients with genotype 1 yielded SVR rates of 80%, around 90% of these patients were eligible for truncated therapy of 24 weeks in a response guided treatment

setting [47] [48]. Very similar results were reported for patients with prior relapse in the PROMISE trial [49]. In the ATTAIN study 771 treatment-experienced partial and null-responder patients were randomized to either simeprevir plus pegIFN and RBV or telaprevir plus pegIFN and RBV. Although efficacy rates were similar (SVR was 55% and 54%, respectively) the safety profile of simeprevir was significantly improved, in particular with regards to anemia (13% vs. 37%) and pruritus (31% vs. 43%), while serious adverse events (SAEs) were reported by 2% and 9% of patients, respectively [50]. Notably, among patients infected with HCV genotype 1a the presence of a common Q80K polymorphism (pre-existing resistance-associated variant or not) results in significantly reduced response rates and thus, it is recommended that patients infected with HCV genotype 1a are screened for this mutation, and if the respective variant is present, consideration is given to selecting an alternative therapy [51].

Sofosbuvir acts as an RNA chain terminator within the catalytic site of the NS5B polymerase. It was approved by the FDA in December 2013 and by the EMA in January 2014 for treatment of genotype 1, 4, 5, and 6 along with pegIFN plus RBV and in genotype 2 and 3 patients as an interferon-free regimen with RBV only.

In the NEUTRINO phase III trial with sofosbuvir plus pegIFN/RBV in 326 treatment-naïve genotype 1, 4, 5 and 6 patients, the overall SVR was 90% (92% in genotype 1a and 82% in genotype 1b; 80% in cirrhotic patients) with a tolerability profile similar to pegIFN plus RBV. One further advantage of this triple treatment regimen is the treatment duration of just 12 weeks [52].

Data on the interferon-free combination of sofosbuvir plus RBV in treatment-naïve patients with genotype 1 are only available from small trials and results are somewhat inconsistent. When given for a duration of 24 weeks SVR rates of 50-68% have been reported and this regimen is currently only recommended for patients who cannot take pegIFN [45] [46] [53] [54].

Thus, currently available approved treatment regimens are not optimal for many patients and there is a clear unmet need for effective anti-HCV compounds which can increase the likelihood of successful treatment and/or decrease the need for pegIFN as components of CHC therapy, ideally with shorter treatment duration.

Combinations of multiple DAAs targeting different steps of viral replication have the potential to significantly improve CHC treatment compared to current therapies by increasing SVR rates, eliminating interferon as a component of therapy, increasing the safety and tolerability of treatment, shortening duration of therapy and simplifying the treatment algorithm. In addition, wider application of DAA therapy and better responses

with combination DAA regimens could significantly reduce the public health burden of this disease.

AbbVie's interferon-free regimen for the treatment of CHC includes 3 DAAs targeting different steps in HCV replication. Paritaprevir (ABT-450) is a NS3/4A protease inhibitor with nanomolar potency *in vitro* and is co-administered with low-dose ritonavir, an inhibitor of the cytochrome P-450 enzyme CYP3A4. As a pharmacologic enhancer of paritaprevir, ritonavir co-administration with paritaprevir (paritaprevir/r) results in higher drug exposures than administration of paritaprevir alone [55]. Ombitasvir (ABT-267) is a nonstructural protein 5A (NS5A) inhibitor with picomolar potency *in vitro*, and dasabuvir (ABT-333) is a NS5B non-nucleoside polymerase inhibitor with nanomolar potency *in vitro*.

The 3 DAA combination of paritaprevir/r – ombitasvir plus dasabuvir with or without RBV has been initially evaluated in 6 Phase III studies with genotype 1 infected patients (SAPPHIRE-I [56], SAPPHIRE-II [57], PEARL-II [58], PEARL-III [59], PEARL-IV [59], TURQUOISE-II [60]).

Therapy for 12 weeks with the above regimen in non-cirrhotic patients resulted in the following SVR rates 12 weeks after EoT (SVR12):

| Table 1 | - SVR12 | rates in | clinical | trials: |
|---------|---------|----------|----------|---------|
|---------|---------|----------|----------|---------|

| Population and treatment duration | Genotype | SVR12<br>ABBVIE REGIMEN + RBV | SVR12<br>ABBVIE REGIMEN alone |
|---|---|---|---|
| treatment duration | | ABBVIE REGIMEN : RBV | ABBVIE REGIMEN alone |
| Non-cirrhotic, | 1a | 95-97% | 90% |
| treatment-naïve (12 weeks) | | (SAPPHIRE-I, PEARL-IV) | (PEARL-IV) |
| (12 Weeks) | 1b | 98-99.5% | 99% |
| | | (SAPPHIRE-I, PEARL-III) | (PEARL-III) |
| Non-cirrhotic, | 1a | 96% | n.a. |
| treatment-<br>experienced | | (SAPPHIRE-II) | |
| (12 weeks) | 1b | 97% | 100% |
| (12 WGGNS) | | (SAPPHIRE-II, PEARL-II) | (PEARL-II) |

These results suggest that the ABBVIE REGIMEN with RBV is the optimal regimen for genotype 1a infected patients, while patients with genotype 1b do not require RBV.

The TURQUOISE-II [60] study explored the efficacy of the ABBVIE REGIMEN in the traditionally most difficult-to-treat cirrhotic patients. This large study enrolled exclusively



genotype 1 infected patients with cirrhosis, including treatment-naïve and treatmentexperienced individuals. All patients received the ABBVIE REGIMEN with RBV and were randomized to 12 or 24 weeks of therapy. Overall 92% and 96% of patients achieved SVR following treatment for 12 or 24 weeks, respectively. Analysis of subgroups demonstrated that the small difference in SVR between treatment arms was due largely to the subgroup of genotype 1a treatment-experienced prior null responders treated for 12 weeks who achieved an SVR of 80%. This subgroup of patients achieved an SVR of 93% when treated for 24 weeks. Among genotype 1a infected patients, partial responders and relapsers had higher SVR rates than null responders in the 12 week treatment group, while similar SVR rates were seen among the null responders, partial responders and relapsers treated for 24 weeks, suggesting that the longer duration of 24 weeks is required only for cirrhotic genotype 1a null responders. SVR rates were very high across all subgroups in genotype 1b treatment-experienced patients treated for 12 and 24 weeks.

The ABBVIE REGIMEN has been studied with and without RBV in over 2,300 patients in Phase III trials across a variety of patient populations including those with compensated cirrhosis. Based on Phase III data, the ABBVIE REGIMEN, with or without RBV, was well tolerated with a low discontinuation rate. Adverse events (AEs) were typically mild, and many of the AEs and laboratory abnormalities reported were attributable to the presence of RBV. However, these AEs were much milder than observed when RBV was given in combination with interferon. Transient, asymptomatic serum alanine aminotransferase (ALT) elevations were observed at a low rate, were not associated with hepatic dysfunction and generally resolved with ongoing treatment. A disproportionate number of the cases were in women on concurrent ethinyl estradiol-containing therapy (i.e., contraceptives or hormone replacement) and discontinuation of the hormonal therapy with continuation or brief interruption of the ABBVIE REGIMEN led to resolution in serum ALT elevation. Transient elevations in serum bilirubin (predominantly indirect) were observed in subjects receiving the ABBVIE REGIMEN with RBV, related to the inhibition of the bilirubin transporters, organic anion-transporting polypeptides (OATPs) 1B1/1B3, by paritaprevir and RBV-induced hemolysis. Bilirubin elevations occurred after initiation of treatment, peaked by study Week 1, and generally resolved with ongoing therapy. Bilirubin elevations were not associated with aminotransferase elevations. The frequency of indirect bilirubin elevations was lower among subjects who did not receive RBV.

Response of CHC genotype 4 was assessed in the phase II study PEARL-I in which 86 treatment-naīve patients were randomized to the 2 DAA combination of Paritaprevir/r ombitasvir with vs. without RBV for 12 weeks. The SVR was 100% with RBV vs. 91% without RBV [61]. No serious SAEs or AEs leading to discontinuation were reported.

These results from pivotal studies are encouraging and the new interferon-free regimens might provide physicians with the armamentarium to cure the vast majority of patients infected with CHC. However, the medical community is expecting data which show how these results translate into routine clinical practice particularly after the experience with the first protease inhibitors which were available to physicians and where the outcome in everyday life and especially the tolerability was far less favorable in certain difficult-to-treat patient subgroups than expected from the development trials [62] [63].

### 7.2 Rationale

The ABBVIE REGIMEN ± RBV for the treatment of CHC has been shown to be safe and effective in randomized controlled clinical trials with strict inclusion and exclusion criteria under well controlled conditions.

The ABBVIE REGIMEN is available in Israel for the treatment of CHC since 2015.

The rationale for this observational study is to determine how the efficacy and safety of the ABBVIE REGIMEN as demonstrated in pivotal trials translates into real world everyday clinical settings, evaluating its effectiveness. Whereas efficacy can be defined as a measure of the capacity of a treatment to produce the desired effect in a controlled environment, such as in a randomized controlled trial, effectiveness is 'the extent to which a drug achieves its intended effect in the usual clinical setting' [64]. Effectiveness trials typically have limited exclusion criteria and will involve the broader patient populations in routine clinical practice, treated per local label, which might include patients with heterogenous compliance patterns and patients with significant comorbid conditions and could be used to model and disseminate best practices. Effectiveness research allows for external patient-, provider-, and system-level factors and can therefore be relevant for health-care decisions by both providers in practice and policy-makers [65].

This observational study is the first effectiveness research examining the ABBVIE REGIMEN ± RBV, used according to local label, under real world conditions in Israel in clinical practice patient population.

During the last decade when dual therapy with pegIFN plus RBV was standard of care for the treatment of CHC, management of patients and clinical outcome were improved following the discovery of predictive factors of virological response, often in observational studies with large data bases [66]. Thus treatment could be targeted to patients most likely to respond and futile treatment stopped in patients with a low likelihood of virological cure. HCV genotype and subtype, baseline viral load, fibrosis stage, age, treatment exposure and on-treatment virological response proved to be useful predictors

for the eradication of HCV in everyday clinical practice [27]. More recently the discovery of a genetic disposition of the Interleukin 28B (IL28B) single nucleotide polymorphism (SNP) contributed further to our understanding of virological responses to treatment [67]. For new interferon-free treatment regimens knowledge of predictive factors of virological response is extremely sparse and several of the now well established predictors of response were not initially identified through analyses of the development trials. This observational study may play an important part in bridging the data gaps and could help identify predictive factors of virological response in everyday clinical settings which were not detected in interventional trials and which could be used to further optimize treatment with the interferon-free ABBVIE REGIMEN in the future.

The label of the ABBVIE REGIMEN will vary according to HCV genotype/subtype and stage of liver disease. It is therefore relevant to understand the pattern of use and outcome in daily clinical practice. In addition, this study will provide data on the impact of adherence on treatment outcomes in everyday settings, which may help treating physicians to improve the management of patients under their care.

The aim of this observational study is to provide evidence of the effectiveness of the interferon-free regimen of Paritaprevir/r – Ombitasvir, ± Dasabuvir, ± Ribavirin and Patient Support Program and its influence on patients with CHC in a real world setting across clinical practice patient populations.

## 8.0 Research Question and Objectives

#### 8.1 Research Question

What is the effectiveness of the interferon-free regimen of Paritaprevir/r – Ombitasvir, ± Dasabuvir, ± Ribavirin and PSP and its influence on patients with CHC in a real life setting across clinical practice patient populations?

### 8.2 Objectives

### 8.2.1 Primary Objective

1. To describe in routine clinical practice the effectiveness of the interferon-free ABBVIE REGIMEN ± RBV in patients with CHC as evidenced by SVR12

### 8.2.2 Secondary Objectives

- 2. To provide real world evidence for predictive factors of virological response
- 3. To describe the pattern of real world use of the ABBVIE REGIMEN ± RBV with respect to different patient and treatment characteristics
- 4. To evaluate the contribution of the patient support program (PSP) to disease control, treatment continuation over time, patient satisfaction and PSP utilization
- 5. To describe the effect of the ABBVIE REGIMEN ± RBV on metabolic profile
- 6. To evaluate the effect of the ABBVIE REGIMEN ± RBV on extrahepatic manifestations and associated diseases like cryoglobulinemia/cutaneous vasculitis or porphyria cutanea tarda

### 9.0 Research Methods

### 9.1 Study Design

This is a prospective, multi-center observational study in patients receiving the interferonfree ABBVIE REGIMEN with or without RBV. The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice and label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.

Adult patients chronically infected with HCV, receiving the interferon-free ABBVIE REGIMEN will be offered the opportunity to participate in this study during a routine clinical visit at the participating sites.

After written informed consent has been obtained, patient data including demographic data, HCV disease characteristics, co-morbidities, co-medication, treatment details, and laboratory assessments as recorded in the patient's medical records (source documentation) will be documented in the electronic case report form (eCRF). Patients will be observed for the duration of the ABBVIE REGIMEN therapy and for up to 24 weeks after treatment completion. No patient identifiable information will be captured, a unique patient number will be automatically allocated by the web based eCRF system once the investigator or designee creates a new patient file.

This study is focusing on collecting real-world data. Follow-up visits, treatment, procedures and diagnostic methods will follow physicians' routine clinical practice. The observational study period entails the following data collection schemes, data documented will be those closest to the time windows as indicated in Figure 1:

- 12-week treatment regimen: four visits plus two interim data collection windows
- 24-week treatment regimen: four visits plus three interim data collection windows

This schedule is based on the anticipated regular follow-up for patients undergoing treatment for CHC.

Figure 1 - Study Flowchart



### 9.2 Setting

For overall research design and observational documentation schedule refer to Sections 9.1 and 9.4.1 as well as to Figure 1.

### 9.2.1 Target Population

Patients are eligible for observation in this cohort if the following applies:

- Treatment-naïve or -experienced adult male or female patients with confirmed CHC, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV according to standard of care and in line with the current local label
- If RBV is co-administered with the ABBVIE REGIMEN, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy)

- Patients must voluntarily sign and date an informed consent form prior to inclusion into the study
- Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial

### 9.2.2 Study Duration

This is a prospective, observational study. The inclusion period will be approximately 8 months and the observational period of the study will be from baseline visit until 24 weeks post-treatment.

The observational period for patients receiving 12 weeks of ABBVIE REGIMEN will be max. 36 weeks (12 weeks treatment and 24 weeks post-treatment observation) and for patients receiving 24 weeks of ABBVIE REGIMEN the observational period will be max. 48 weeks (24 weeks treatment and 24 weeks post-treatment observation).

#### 9.2.3 Termination Criteria

For patients who terminate the ABBVIE REGIMEN prematurely for whatever reason the EoT eCRF page should be filled in and the reason for treatment discontinuation should be documented. If the reason for ABBVIE REGIMEN discontinuation is due to an SAE, the event must be reported to AbbVie within 24 hours of physician awareness (see Section 11.1.5).

If, in such patients, there is evidence of virological response during therapy or at EoT, the SVR12 and SVR24 pages should be completed if respective data is available.

### 9.2.4 Investigator Selection Criteria

Medical centers and outpatient clinics qualified by training and experience in the management of patients with CHC will be selected to participate in this study. The AbbVie Affiliate Medical Director will ensure that sites participating in the study are representative of the medical practice in the country, have the ability to conduct the study and their availability of the target patient population. The type of the participating treating institute will be documented in the eCRF.

### 9.3 Variables

### 9.3.1 Primary Variable

 The percentage of patients achieving SVR12 (HCV RNA <50 IU/mL 12 weeks [i.e. ≥70 days] after the last actual dose of the ABBVIE REGIMEN)

### 9.3.2 Secondary Variables

- Type of treatment regimen (± Dasabuvir, ± RBV, intended and actual combination, dose and duration)
- PAM-13, PSP satisfaction and utilization questionnaires
- Metabolic laboratory profile (see section 9.4.1.1) prior to treatment initiation, and at all subsequent visits
- Cryoglobulins, immunoglobulins and porphyrin prior to treatment initiation, and at all subsequent visits

#### 9.4 Data Sources

Source documents are defined as original documents. The investigator will document patient data in his/her own patient files which will serve as source data for the study. Data are collected from the source documents for each patient in the study, consisting of medical records containing demographic data, medical, treatment and diagnostic documentation and laboratory assessments.

The investigator(s)/institution(s) will permit study-related monitoring, audits, independent ethics committee/- review board (IEC/IRB) review, and regulatory inspection(s), providing direct access to source data documents.

#### 9.4.1 Data to be Documented

This observational study covers three documentation periods, see Figure 1. An overview on data to be collected throughout the study is summarized in **Table 2**.

After the patient has signed the informed consent form, the following data will be documented in the eCRF, if available from the patient charts based on assessments done in physicians' routine clinical practice.

### 9.4.1.1 Inclusion Documentation

The following will be documented:

- Demographic information
  - o Interleukin 28B (IL28B) genotypes
- CHC disease characteristics
  - Year of diagnosis and mode of infection
  - Stage of liver fibrosis
- CHC treatment history
  - Naïve or experienced
  - o If experienced, most recent prior therapy and outcome
- Relevant medical history, co-morbidities and co-infections
- Concomitant medication, see 9.4.1.5
- ABBVIE REGIMEN ± RBV
- Laboratory data

| aboratory data | |
|---|---|
| Key clinical chemistry | Remarks |
| <ul><li>ALT</li></ul> | including upper limit of normal (ULN), |
| (alanine-aminotransferase) | |
| <ul><li>AST</li></ul> | including ULN, |
| (aspartate-aminotransferase) | AST to platelet ratio index (APRI) and Fibrosis-4 Score/Index (FIB-4)* will be calculated |
| <ul><li>y-GT</li></ul> | |
| (gamma-glutamyltransferase) | |
| <ul><li>Total bilirubin</li></ul> | |
| <ul><li>Albumin</li></ul> | |
| <ul><li>Creatinine</li></ul> | creatinine clearance <sup>#</sup> will be calculated |

### Key hematology

AFP

- Hb (Hemoglobin)
- Platelets
- Prothrombin time or international normalized ratio (INR)

#### Virology

- HCV genotype and subtype
- HCV RNA quantitative/ qualitative HCV RNA by polymerase chain reaction (PCR) test, see 9.4.1.4

#### HIV-infected patients only

- CD 4 count most recent assessment (cluster of differentiation 4)
- HIV RNA in copies/mL

\*by Cockcroft-Gault-Formula based on creatinine, gender, age and weight

 Metabolic profile: Fasting glucose, fasting insulin (HOMA score will be calculated by eCRF based on fasting insulin and glucose), HbA1c, fasting high-density

<sup>\*</sup>derived from patient's age, ALT, AST and platelets

- lipoprotein (HDL), fasting low-density lipoprotein (LDL), fasting cholesterol and fasting triglycerides
- More extensive laboratory: direct bilirubin, indirect bilirubin, AFP, Fibrotest, cryoglobulin presence, cryocrit, IgG, IgA, IgM, rheumatoid factor (RF), complement components, proteinuria, microscopic hematuria, cutaneous vasculitis score, plasma and urinary porphyrin, ferritin, drug monitoring of calcineurin (CNI) inhibitors (for OLT patients only)
- PAM-13

### 9.4.1.2 During Treatment Documentation

Follow-up visits are scheduled by the physician per routine clinical practice. Likewise treatment, procedures and diagnostic methods will follow physicians' routine clinical practice.

The following will be documented:

Laboratory data

| Key clinical chemistry | <u>Remarks</u> |
|------------------------|-----------------------------------|
| <ul><li>ALT</li></ul> | including ULN |
| <ul><li>AST</li></ul> | including ULN, |
| | APRI and FIB-4 will be calculated |

γ-GT

Total bilirubin

Creatinine clearance will be calculated

#### Key hematology

Hb

Platelets

#### Virology

HCV RNA quantitative/ qualitative HCV RNA PCR test, see 9.4.1.4

### HIV-infected patients only

CD 4 count most recent assessment

HIV RNA in copies/mL

- Concomitant medication, see 9.4.1.5
- Adherence to ABBVIE REGIMEN ± RBV (ABBVIE REGIMEN % of target dose taken and RBV Y/N)
- Tolerability (sAEs and AEs, see 11.1.5) and pregnancies (see 11.1.6)
- Metabolic profile: Fasting glucose, fasting insulin (HOMA score will be calculated by eCRF based on fasting insulin and glucose), HbA1c, HDL, LDL, fasting cholesterol and fasting triglycerides
- More extensive laboratory: direct bilirubin, indirect bilirubin, AFP, Fibrotest, cryoglobulin presence, cryocrit, IgG, IgA, IgM, RF, complement components, proteinuria, microscopic hematuria, cutaneous vasculitis score, plasma and urinary porphyrin, ferritin, drug monitoring of CNI inhibitors (for OLT patients only)

PSP satisfaction and utilization questionnaires; PAM-13

### 9.4.1.3 Post-Treatment Documentation

Follow-up visits are scheduled by the physician per routine clinical practice. Likewise treatment, procedures and diagnostic methods will follow physicians' routine clinical practice.

The following will be documented:

Laboratory data

| Key clinical chemistry | <u>Remarks</u> |
|------------------------|------------------------------------|
| <ul><li>ALT</li></ul> | including ULN |
| <ul><li>AST</li></ul> | including ULN, |
| | APRI and FIB-4, will be calculated |

γ-GT

Total bilirubin

AlbuminCreatinine

Creatinine clearance will be calculated

#### Key hematology

Hb

Platelets

Prothrombin time or INR

#### Virology

HCV RNA quantitative/ qualitative HCV RNA PCR test, see 9.4.1.4

#### HIV-infected patients only

CD 4 count most recent assessment

HIV RNA in copies/mL

- Tolerability (sAEs, see 11.1.4) and pregnancies (see 11.1.6)
- Metabolic profile: Fasting glucose, fasting insulin (HOMA score will be calculated by eCRF based on fasting insulin and glucose), HbA1c, HDL, LDL, fasting cholesterol and fasting triglycerides
- More extensive laboratory: direct bilirubin, indirect bilirubin, AFP, Fibrotest, cryoglobulin presence, cryocrit, IgG, IgA, IgM, RF, complement components, proteinuria, microscopic hematuria, cutaneous vasculitis score, plasma and urinary porphyrin, ferritin, drug monitoring of CNI inhibitors (for OLT patients only)
- PSP Satisfaction and utilization questionnaires

Table 2 - Data Documentation Schedule

| Assessment/ Procedure | 0 | Treat | ment Period | ł | Post-tr | eatme<br>Period | |
|---|---|---|---|---|---|---|---|
| (only available data to be collected; no diagnostic or monitoring procedures to be applied to the patients apart from those of routine clinical practice) | Baseline | On-<br>treatment<br>visits | Mid<br>treatment<br>visit for pts<br>receiving<br>24 weeks<br>of therapy | EoT <sup>b</sup> | Early<br>PT visit | SVR<br>12<br>visit | SVR<br>24<br>visit |
| Patient Informed Consent | Xa | | | | | | |
| Demographic information | X | | | | | | |
| IL28B | Х | | | | | | |
| Relevant CHC disease characteristics | X | | | | | | |
| Liver fibrosis stage | X | | | | | | |
| CHC treatment history | X | | | | | | |
| HCV genotype and subtype | X | | | | | | |
| HCV RNA samples | X | Χ | Х | Х | Х | X | X |
| Clinical chemistry and hematology | X | Х | X | X | Х | X | X |
| ABBVIE REGIMEN initiation documentation | X | | | | | | |
| ABBVIE REGIMEN adherence | | Х | Х | Х | | | |
| Concomitant medication | X | Х | X | Х | | | |
| Relevant medical history, co-morbidities | X | | | | | | |
| sAE, AE and pregnancy reporting | X | Х | Χ | Х | Xc | $X_q$ | $X_q$ |
| For patients receiving RBV: Evidence, in accordance with local label, that female patient or female partner of male patient is not pregnant | X | 0.000 | | | | | |
| Metabolic profile | X | X | X | X | X | X | X |
| Additional laboratory assessments | X | Х | Х | Χ | Х | X | X |
| Patient questionnaire - PAM-13 | X | | | Χ | 5 | | |
| PSP evaluation | 5 | X | X | Х | Х | X | |

Abbreviations: EoT = End of Treatment (at Week 12 or 24 or at premature discontinuation), PT = Post-Treatment

- a Written informed consent must be obtained before any data documentation in the eCRF
- b Patients who prematurely discontinue should return to the site to document EoT data
- c Tolerability documentation until PT week 4
- d Pregnancy reporting for patients treated with DAA plus RBV

### 9.4.1.4 HCV RNA Sample

**HCV RNA sample** – the following needs to be documented:

- Quantitative HCV RNA by PCR test
  - o Test name and result in IU/mL

Confidential Information

- Lower limit of detection (LLoD) in IU/mL and lower limit of quantification (LLoQ) in IU/mL
- Qualitative HCV RNA by PCR test
  - Test name and result (positive/negative)
  - o LLoD in IU/mL

#### 9.4.1.5 Concomitant Medication

Concomitant medication - the following will be documented:

 Concomitant medication used from the time when the decision is made to initiate treatment with the ABBVIE REGIMEN until after the last dose

It should be verified by the treating physician that concomitant medication can be safely administered with the ABBVIE REGIMEN (including ritonavir) and RBV. Some medications may be contra-indicated, some may require dose adjustments due to potential for drug-drug interactions (DDIs). The investigator or qualified designee should review the concomitant medication(s) labels and screen concomitant medications at each visit for potential DDIs.

### 9.4.1.6 Standardized Assessment Tools

#### Patient Activation Measure – (PAM-13)

PAM 13 is a measure used to assess the patient knowledge, skill, and confidence for self-management. It should require approximately 7 minutes to complete and is presented in Annex 3.

### Patient Support Program (PSP) Questionnaire

The PSP utilization and satisfaction assessment will evaluate the frequency of utilization and patient's overall satisfaction with their respective Patient Support Program.

The PSP questionnaire should require approximately 2-5 minutes to complete and is presented in Annex 5-6.

### 9.5 Study Size

In phase III studies investigating the interferon-free ABBVIE REGIMEN  $\pm$  RBV, SVR12 rates of at least 90% were observed, even in difficult-to-treat CHC patients (e.g. cirrhotic G1a treatment experienced patients). To describe in routine clinical practice the effectiveness of the ABBVIE REGIMEN  $\pm$  RBV in patients with CHC, a precise estimate of the SVR12 rates should be achieved.

It is expected, that during the planned inclusion period of 8 months about 250 patients treated with the ABBVIE REGIMEN ± RBV can be included. It is furthermore, expected, that the number of patients to exclude from the core population will be not higher than 5-10%. With 235 evaluable patients the width of the 95% confidence interval (CI) will be 7.7% and 5.7% for SVR12 rates of 90% and 95%, respectively. If only 200 patients can be evaluated, the 95% CI will have a width of less than 8.4% for a SVR12 rate of at least 90% and less than 6.2% for a SVR12 rate of at least 95%. See for further details.

| Table 3- Width of 95% Confidence Interval for SV | /R1 | ₹′ | 1 | ı | i | ì | ì | 2 | i | | | ı | ı | ı | ı | 1 | 1 | 1 | 1 | 1 | 1 | 7 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | ı | ξ | ţ | ۹ | ł | ı | ı | ı | 1 | ٧ | ١ | ١ | ľ | ì | ۶ | ٥ | 2 | 3 | 3 | ٥ | Č | ٤ | ì | ì | ì | ì | ÷ | , | | | | | • | r | r | 1 | ı١ | ) | 0 | ĺ | ( | ľ | ľ | Ī | 1 | 1 | | | | ı | ı | ı | 1 | 3 | ć | ć | 7 | V | ١ | 7 | r | ı | ļ | ) | e | E | ľ | 1 | ۱ | ١ | r | ı | | • | е | | C | ( | I | ١ | n | ì | ę | е | Е | 1 | O | C | ľ | ı | П | T | ľ | 1 | ٦ | r | ı | ) | ) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| K | 1 | ĺ | 1 | į | ı | ı | ı | ı | ı | l | ı | Į | | | ļ | ļ | 1 | 1 | 1 | 1 | 1 | 7 | 7 | 7 | 7 | 7 | 1 | 1 | 1 | 1 | Ľ | ζ. | €. | 1 | 7 | 7 | K | K | /K | /K | VK' | VK' | VK. | VK. | VK | VK | VK | )VK | VK | אענ | )VK | >VK | <b>VK</b> | >VK | SVK' | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | )r | <b>3r 5v</b> R | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | TOR SVK | TOR SVK | tor SVK | tor SVK | TOR SVK | I TOR SVK | I TOR SVK | II TOR SVK | II for SVK | al for SVR | ai for SVK | al for SVR | al for SVK | vai for SVK | val for SVR | rval for SVK | rvai for SVR | rval for 5VK | erval for SVK | erval for SVK | erval for 5VK | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for 5VK | interval for SVR | e interval for SVR | e interval for 5vK | ce interval for 5 v K | ce interval for 5 v K | ce interval for 5 v R | ice interval for 5 v K | ice interval for SVR | nce interval for SVR | ence interval for 5 vR | ence interval for SVR | ence interval for 5vR | ence interval for 5 vR | ience interval for SVR | dence interval for 5 vR | dence interval for 5 vR | idence interval for 5 vR | idence interval for 5 vR | ndence interval for 5 vR | fidence interval for 5 vR | Tidence interval for 5 vR | ifidence interval for 5 vR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for 5VR |
| K | 1 | | 1 | | ı | ı | l | ı | l | ı | Į | ı | | | ı | | 1 | 1 | 1 | 1 | 1 | 7 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | Ľ | ζ. | €. | ₹. | 7 | 7 | K | K | /K | /K | VK. | VK' | VK. | VK. | VK. | VK | VK | VK | VK' | VK | <b>VK</b> | <b>VK</b> | SVK' | 3VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | or SVR | or SVR | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | I for SVR | II TOR SVR | II for SVK | al for SVK | ai for SVR | al for SVR | al for SVR | val for SVR | val for SVR | rval for SVR | rval for SVR | rval for SVR | erval for SVR | erval for SVR | erval for SVR | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for SVR | interval for SVR | e interval for SVR | e interval for SVR | ce interval for SVR | ce interval for SVR | ce interval for SVR | ice interval for SVR | nce interval for SVR | nce interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ience interval for SVR | dence interval for SVR | dence interval for SVR | idence interval for SVR | idence interval for SVR | ridence interval for SVR | fidence interval for SVR | fidence interval for SVR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for SVR |
| K | 1 | | 1 | | ı | ı | l | ı | l | ı | Į | ı | | | ı | | 1 | 1 | 1 | 1 | 1 | 7 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | Ľ | ζ. | €. | ₹. | 7 | 7 | K | K | /K | /K | VK. | VK' | VK. | VK. | VK. | VK | VK | VK | VK' | VK | <b>VK</b> | <b>VK</b> | SVK' | 3VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | or SVR | or SVR | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | I for SVR | II TOR SVR | II for SVK | al for SVK | ai for SVR | al for SVR | al for SVR | val for SVR | val for SVR | rval for SVR | rval for SVR | rval for SVR | erval for SVR | erval for SVR | erval for SVR | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for SVR | interval for SVR | e interval for SVR | e interval for SVR | ce interval for SVR | ce interval for SVR | ce interval for SVR | ice interval for SVR | nce interval for SVR | nce interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ience interval for SVR | dence interval for SVR | dence interval for SVR | idence interval for SVR | idence interval for SVR | ridence interval for SVR | fidence interval for SVR | fidence interval for SVR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for SVR |
| K | 1 | | 1 | | ı | ı | l | ı | l | ı | Į | ı | | | ı | | 1 | 1 | 1 | 1 | 1 | 7 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | Ľ | ζ. | €. | ₹. | 7 | 7 | K | K | /K | /K | VK. | VK' | VK. | VK. | VK. | VK | VK | VK | VK' | VK | <b>VK</b> | <b>VK</b> | SVK' | 3VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | or SVR | or SVR | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | I for SVR | II TOR SVR | II for SVK | al for SVK | ai for SVR | al for SVR | al for SVR | val for SVR | val for SVR | rval for SVR | rval for SVR | rval for SVR | erval for SVR | erval for SVR | erval for SVR | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for SVR | interval for SVR | e interval for SVR | e interval for SVR | ce interval for SVR | ce interval for SVR | ce interval for SVR | ice interval for SVR | nce interval for SVR | nce interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ience interval for SVR | dence interval for SVR | dence interval for SVR | idence interval for SVR | idence interval for SVR | ridence interval for SVR | fidence interval for SVR | fidence interval for SVR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for SVR |
| K | 1 | | 7 | ı | l | ı | ı | ı | ı | ı | Į | Į | | | ļ | ļ | 1 | 1 | 1 | 1 | 1 | 7 | 7 | 7 | 7 | 7 | 1 | 1 | 1 | 1 | Ľ | ζ. | €. | ₹. | 7 | 7 | K | K | /K | /K | VK. | VK' | VK. | VK. | VK. | VK | VK | VK | VK' | VK | <b>VK</b> | <b>VK</b> | SVK' | 3VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | or SVR | or SVR | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | I for SVR | II TOR SVR | II for SVK | al for SVK | ai for SVR | al for SVR | al for SVR | val for SVR | val for SVR | rval for SVR | rval for SVR | rval for SVR | erval for SVR | erval for SVR | erval for SVR | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for SVR | interval for SVR | e interval for SVR | e interval for SVR | ce interval for SVR | ce interval for SVR | ce interval for SVR | ice interval for SVR | nce interval for SVR | nce interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ience interval for SVR | dence interval for SVR | dence interval for SVR | idence interval for SVR | idence interval for SVR | ridence interval for SVR | fidence interval for SVR | fidence interval for SVR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for SVR |
| K | 1 | | 1 | | ı | ı | l | ı | l | ı | Į | ı | | | ı | | 1 | 1 | 1 | 1 | 1 | 7 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | Ľ | ζ. | €. | ₹. | 7 | 7 | K | K | /K | /K | VK. | VK' | VK. | VK. | VK. | VK | VK | VK | VK' | VK | <b>VK</b> | <b>VK</b> | SVK' | 3VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | or SVR | or SVR | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | I for SVR | II TOR SVR | II for SVK | al for SVK | ai for SVR | al for SVR | al for SVR | val for SVR | val for SVR | rval for SVR | rval for SVR | rval for SVR | erval for SVR | erval for SVR | erval for SVR | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for SVR | interval for SVR | e interval for SVR | e interval for SVR | ce interval for SVR | ce interval for SVR | ce interval for SVR | ice interval for SVR | nce interval for SVR | nce interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ience interval for SVR | dence interval for SVR | dence interval for SVR | idence interval for SVR | idence interval for SVR | ridence interval for SVR | fidence interval for SVR | fidence interval for SVR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for SVR |
| K | 1 | | 1 | | ı | ı | l | ı | l | ı | Į | ı | | | ı | | 1 | 1 | 1 | 1 | 1 | 7 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | Ľ | ζ. | €. | ₹. | 7 | 7 | K | K | /K | /K | VK. | VK' | VK. | VK. | VK. | VK | VK | VK | VK' | VK | <b>VK</b> | <b>VK</b> | SVK' | 3VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | or SVR | or SVR | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | I for SVR | II TOR SVR | II for SVK | al for SVK | ai for SVR | al for SVR | al for SVR | val for SVR | val for SVR | rval for SVR | rval for SVR | rval for SVR | erval for SVR | erval for SVR | erval for SVR | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for SVR | interval for SVR | e interval for SVR | e interval for SVR | ce interval for SVR | ce interval for SVR | ce interval for SVR | ice interval for SVR | nce interval for SVR | nce interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ience interval for SVR | dence interval for SVR | dence interval for SVR | idence interval for SVR | idence interval for SVR | ridence interval for SVR | fidence interval for SVR | fidence interval for SVR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for SVR |
| K | | | 1 | | ı | ı | ı | ı | ı | ı | Į | Į | | | ı | | | | | | | 7 | 1 | 1 | 1 | 1 | | | | | Ľ | ζ. | €. | 1 | 7 | 7 | K | K | /K | /K | VK' | VK' | VK. | VK. | VK | VK | VK | )VK | VK | אענ | )VK | >VK | <b>VK</b> | >VK | SVK' | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | )r | <b>3r 5v</b> R | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | TOR SVK | TOR SVK | tor SVK | tor SVK | TOR SVK | I TOR SVK | I TOR SVK | II TOR SVK | II for SVK | al for SVR | ai for SVK | al for SVR | al for SVK | vai for SVK | val for SVR | rval for SVK | rvai for SVR | rval for 5VK | erval for SVK | erval for SVK | erval for 5VK | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for 5VK | interval for SVR | e interval for SVR | e interval for 5vK | ce interval for 5 v K | ce interval for 5 v K | ce interval for 5 v R | ice interval for 5 v K | ice interval for SVR | nce interval for SVR | ence interval for 5 vR | ence interval for SVR | ence interval for 5vR | ence interval for 5 vR | ience interval for SVR | dence interval for 5 vR | dence interval for 5 vR | idence interval for 5 vR | idence interval for 5 vR | ndence interval for 5 vR | fidence interval for 5 vR | Tidence interval for 5 vR | ifidence interval for 5 vR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for 5VR |
| K | | | 1 | | ı | ı | ı | ı | ı | ı | Į | Į | | | ı | | | | | | | 7 | 1 | 1 | 1 | 1 | | | | | Ľ | ζ. | €. | 1 | 7 | 7 | K | K | /K | /K | VK' | VK' | VK. | VK. | VK | VK | VK | )VK | VK | אענ | )VK | >VK | <b>VK</b> | >VK | SVK' | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | )r | <b>3r 5v</b> R | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | TOR SVK | TOR SVK | tor SVK | tor SVK | TOR SVK | I TOR SVK | I TOR SVK | II TOR SVK | II for SVK | al for SVR | ai for SVK | al for SVR | al for SVK | vai for SVK | val for SVR | rval for SVK | rvai for SVR | rval for 5VK | erval for SVK | erval for SVK | erval for 5VK | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for 5VK | interval for SVR | e interval for SVR | e interval for 5vK | ce interval for 5 v K | ce interval for 5 v K | ce interval for 5 v R | ice interval for 5 v K | ice interval for SVR | nce interval for SVR | ence interval for 5 vR | ence interval for SVR | ence interval for 5vR | ence interval for 5 vR | ience interval for SVR | dence interval for 5 vR | dence interval for 5 vR | idence interval for 5 vR | idence interval for 5 vR | ndence interval for 5 vR | fidence interval for 5 vR | Tidence interval for 5 vR | ifidence interval for 5 vR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for 5VR |
| K | 1 | ĺ | 1 | ļ | ı | ı | ı | ı | ı | l | Į | Į | | | Į | J | | | | | | | 1 | 1 | | | | | | | Ľ | ζ. | €. | 1 | 7 | 7 | K | K | /K | /K | VK' | VK' | VK. | VK. | VK | VK | VK | )VK | VK | אענ | )VK | >VK | <b>VK</b> | >VK | SVK' | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | )r | <b>3r 5v</b> R | or SVK | or SVK | or SVK | or SVK | or SVK | ror SVK | TOR SVK | TOR SVK | tor SVK | tor SVK | TOR SVK | I TOR SVK | I TOR SVK | II TOR SVK | II for SVK | al for SVR | ai for SVK | al for SVR | al for SVK | vai for SVK | val for SVR | rval for SVK | rvai for SVR | rval for 5VK | erval for SVK | erval for SVK | erval for 5VK | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for 5VK | interval for SVR | e interval for SVR | e interval for 5vK | ce interval for 5 v K | ce interval for 5 v K | ce interval for 5 v R | ice interval for 5 v K | ice interval for SVR | nce interval for SVR | ence interval for 5 vR | ence interval for SVR | ence interval for 5vR | ence interval for 5 vR | ience interval for SVR | dence interval for 5 vR | dence interval for 5 vR | idence interval for 5 vR | idence interval for 5 vR | ndence interval for 5 vR | fidence interval for 5 vR | Tidence interval for 5 vR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for 5VR |
| K | 1 | | 1 | ı | ı | ı | ı | ı | ı | ı | ı | ı | ı | Į | | | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | ï | ĺ. | €. | 1 | 7 | 7 | K | K | /K | /K | VK' | VK. | VK | VK | VK | VK | VK | VK | VK | VK | VK | VK | SVK | <b>SVK</b> | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r SVK | or SVK | or SVK | or SVK | or SVK | or SVK | or SVK | or SVK | for SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | tor SVK | I for SVK | II TOR SVK | II for SVK | al for SVK | ai for SVR | al for SVR | al for SVR | val for SVR | val for SVR | rval for SVR | rvai for SVR | rval for SVR | erval for SVR | erval for SVR | erval for SVR | terval for SVR | terval for SVR | iterval for SVR | iterval for SVR | nterval for SVR | interval for SVR | interval for SVR | interval for SVR | e interval for SVR | e interval for SVR | ce interval for SVR | ce interval for SVR | ce interval for SVR | ice interval for SVR | nce interval for SVR | nce interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ence interval for SVR | ience interval for SVR | dence interval for SVR | dence interval for SVR | idence interval for SVR | idence interval for SVR | ridence interval for SVR | fidence interval for SVR | fidence interval for SVR | ifidence interval for SVR | ntidence interval for SVR | nfidence interval for SVR | ntidence interval for SVR |
| K | | | | Į | l | L | I | L | I | l | Į | Į | | | | | | | | | | | | | | | | | | | Ĺ | ٤ | ۲ | ۲ | ヽ | ス | ĸ | K | /K | /K | ٧ĸ | ٧ĸ | ٧ĸ | VK | VK | VK | VK | VK | ٧K | ٧ĸ | ٥VK | ٥VK | vĸ | ٥VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | rsvk | r svk | )r | )r 5 v K | or SVK | or SVK | or 5vk | or SVK | or SVK | ror SVK | tor SVK | TOR SVK | tor SVK | tor SVK | tor SVK | TOF SVK | I TOR SVK | II TOR SVK | II TOR SVK | ai for SVR | ai for SVR | al for SVR | ai for 5vR | vai for SVR | vai for SVR | rvai for SVR | rvai for 5vR | rval for 5VK | erval for 5vK | ervai for SVR | ervai for SVK | terval for 5vK | terval for 5vK | iterval for 5vK | iterval for 5vK | nterval for 5vK | interval for 5vK | interval for 5VK | interval for 5vK | e interval for 5vK | e interval for 5vK | e interval for 5vK | ce interval for 5vK | ce interval for 5vK | ice interval for 5vK | ice interval for 5 v K | nce interval for 5vK | ince interval for 5 v K | ence interval for 5vK | ence interval for 5vK | ence interval for 5vK | ience interval for 5vK | aence interval for 5vK | dence interval for 5vK | idence interval for 5vK | idence interval for 5vK | ndence interval for 5vK | fidence interval for 5vK | maence interval for 5vK | ifidence interval for 5VK | ntidence interval for 5vK | nfidence interval for 5vK | ntidence interval for 5VK |
| K | ď | ď | | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | | | | | | | | | | | | | | | į | ĺ | ζ | < | ヽ | ス | ĸ | K | /K | /K | ٧K | ٧ĸ | ٧ĸ | VK | VK | VK | VK | VK | ٧K | ٧K | ٥VK | ٥VK | >VK | >VK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | rsvk | r Svk | )r | or Svk | or SVK | or SVK | or 5vk | or SVK | or SVK | ror SVK | tor SVK | TOR SVK | tor 2 NK | tor SVK | tor 2 kg | I TOR SVK | I TOR SVK | II TOR SVK | II TOR SVK | ai tor SVK | ai for SVK | al for SVK | ai for SVK | vai for SVR | vai for SVR | rvai for 5vK | rvai for SVK | rval for 5VK | erval for 5vK | erval for 5vK | ervai for 5vK | terval for 5vK | tervai for 5vK | itervai for 5 v K | itervai for SVR | nterval for 5vK | interval for 5vR | interval for 5VK | interval for SVR | e interval for 5vK | e interval for 5vK | e interval for 5vK | ce interval for 5 v R | ce interval for 5 v R | ice interval for 5 v R | ice interval for 5 v K | nce interval for 5 v R | ince interval for 5 v R | ence interval for 5 v R | ence interval for 5vK | ence interval for 5vK | ience interval for 5vK | aence interval for 5vK | dence interval for 5vK | idence interval for 5 v R | idence interval for 5 vR | fidence interval for 5 v R | fidence interval for 5 v R | maence interval for 5vK | ifidence interval for 5 v R | ntidence interval for 5 vR | nfidence interval for 5VR | ntidence interval for 5VK |
| K | ί | ί | | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | ĺ | ĺ | ĺ | ĺ | ĺ | ĺ | ľ | ľ | ľ | ľ | ľ | ĺ | ĺ | ĺ | ĺ | | í | í | 1 | 7 | ٦ | K | K | /K | /K | ٧K | ٧ĸ | VK | VK | VK | VK | VK | VK | VK | ٧ĸ | ) V K | งห | >VK | วงห | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | SVK | r SVK | r Svk | )r | )r 5 v k | or Svk | or 5 v K | or Svk | Or SVK | or SVK | ror SVK | TOR SVK | TOR SVK | tor 2AK | tor 2AK | TOL 2AK | I TOR SVK | I TOL 2AK | II TOR SVK | II TOR SVK | ai for Syk | ai for SVK | al for SVK | ai for Syk | vai for SVK | vai for SVR | rvai for SVK | rvai for SVK | rval for 5vk | erval for 5vk | erval for 5vk | ervai for 5vk | terval for 5vK | tervai for 5 v K | iterval for 5 v K | iterval for 5vk | nterval for 5 v K | interval for 5 v R | interval for 5VK | interval for 5vK | e interval for 5 v R | e interval for 5vK | e interval for 5vK | ce interval for 5vK | ce interval for 5vk | ice interval for 5 v R | ice interval for 5vK | nce interval for 5 v R | ence interval for 5 v R | ence interval for 5 v R | ence interval for 5 v R | ence interval for 5 v R | ience interval for 5 v R | aence interval for 5vk | dence interval for 5 v R | idence interval for 5 v R | idence interval for 5 v R | lidence interval for SVR | fidence interval for 5 v R | maence interval for 5 v R | ifidence interval for SVR | ntidence interval for 5 v R | nfidence interval for 5 v R | ntidence interval for 5VK |
| r | ί | ί | ľ | П | П | .1 | .1 | .1 | .1 | .1 | .1 | .1 | .1 | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | ľ | í | | ١ | 4 | 7 | 7 | r | r | /r | /r | ۷r | ۷r | VF | VF | VF | VF | VF | VF | Vr | Vr | งงห | אטכ | วงห | ンVド | ンVド | SVr | องห | SVr | <b>37</b> F | <b>21</b> 1 | <b>21</b> 1 | SVF | SVF | SVF | SVF | rsvr | rsvr | )r | 2r | or Svr | or Svr | or 5vr | Or SVR | or Syr | ior Syr | tor Svr | TOR SVE | tor 2 A L | TOL 2AL | TOL 2AL | I TOR SVR | I TOR SVR | II TOR SVR | ii tor Svr | ai for Syr | ai for Syr | al for SVR | ai for Syk | vai for Svr | vai for Syr | rvai for Svr | rvai for 5vr | rval for 5vk | erval for 5vr | erval for 5vr | ervai for 5vr | terval for 5vk | terval for 5vr | iterval for 5vk | iterval for 5vk | nterval for 5vk | interval for 5 v R | interval for 5VR | interval for 5vr | e interval for SVR | e interval for 5vr | e interval for 5vr | ce interval for 5vk | ce interval for 5vk | ice interval for 5vr | ice interval for 5vr | nce interval for 5 v R | ence interval for 5vr | ence interval for 5vr | ence interval for 5vr | ence interval for 5vr | ience interval for 5vk | aence interval for 5vk | dence interval for 5vk | idence interval for 5vk | idence interval for 5vk | ndence interval for 5vk | fidence interval for 5 v R | maence interval for 5vk | ifidence interval for 5 v R | ntidence interval for 5 v R | ntidence interval for 5vk | ntidence interval for 5vk |
| | ľ | ١ | < | <b>く</b> 1 | <b>(</b> 1 | <b>(</b> 1 | <b>K</b> 1 | <b>(</b> 1 | <b>K</b> 1 | <b>(</b> 1 | <b>K</b> 1 | <1 | < | < | < | < | < | < | < | < | < | < | < | < | < | < | < | < | < | < | ٩ | | ۰ | Ì | | | ı | | / | / | ۷I | ٧I | VI | VI | VI | ٧I | VI | V | ועכ | ועכ | ועכ | ועכ | SVI | ועכ | SVI | SVI | องเ | SVI | <b>2 V</b> I | 201 | 201 | SVI | 201 | . 2 V I | . 2AI | r Svi | r Svi | or Svi | or Svi | or Svi | or Svi | or Svi | or Svi | or Svi | ror Svi | tor Svi | tor 201 | tor Svi | tor Svi | tor 201 | I TOF SVI | i tor Svi | II TOR SVI | ai tor Svi | ai tor Svi | ai for Svi | al for Svi | aı tor 5vi | vai for Svi | vai for Svi | rvai for Svi | rvai for Svi | rvai for Svi | ervai for 5 vi | ervai for Svi | ervai for Svi | terval for Svi | tervai for Svi | itervai for Svi | itervai for Svi | nterval for Svi | ıntervai tor 5vi | interval for 5vi | interval for Svi | e interval for Svi | e interval for 5vi | e interval for Svi | ce interval for Svi | ce interval for 5vi | ice interval for Svi | ice interval for Svi | nce interval for Svi | ince interval for 5 vi | ence interval for 5 vi | ence interval for 5vi | ence interval for 5vi | ience interval for 5vi | aence interval for 5vi | dence interval for Svi | idence interval for Svi | idence interval for Svi | ndence interval for Svi | fidence interval for Svi | maence interval for Svi | ifidence interval for Svi | nfidence interval for Svi | nfidence interval for Svi | ntidence interval for 5vi |
| I | 1 | r | K | K1 | RΊ | K1 | RΊ | RΊ | RΊ | K1 | K1 | K1 | K1 | K | K' | K | K | K | K | K | K | K | K | K | K | K | K | K | K | K | r | r | ľ | | | | | 1 | Į | Į | ۷ | ٧ | V | V | V | V | V | V | ›۷ | ٥V | <b>5</b> V | ٥٧ | 5 V | <b>5</b> V | <b>5 V</b> | <b>5</b> V | <b>5</b> V | <b>5</b> V | <b>5</b> V | <b>5</b> V | <b>5</b> V | <b>5</b> V | <b>5</b> V | . <b>5</b> v | . 2 A | rsv | r Sv | )r 5 v | or 5 v | or 5 v | or 5 v | or 5 v | or 5 v | or Sv | ror 5 v | tor 5 v | tor 5 v | tor 5 v | tor 2 v | tor 5 v | i tor 5 v | i tor Sv | II TOR SV | ai tor Sv | ai tor 5 v | ai for Sv | al for Sv | aı tor 5v | vai for 5 v | vai for 5 v | rvai for 5 v | rvai for Sv | rvai for 5 v | ervai for 5 v | ervai for 5 v | ervai for 5 v | tervai for 5 v | tervai for 5 v | itervai for 5 v | itervai for 5 v | ntervai for 5 v | ıntervai tor 5 v | interval for 5 v | interval for 5 v | e intervai for 5 v | e interval for 5 v | ce interval for 5 v | ce interval for 5 v | ce interval for 5 v | ice interval for 5 v | ice interval for 5 v | nce interval for 5 v | ence interval for 5 v | ence interval for 5 v | ence interval for 5 v | ence interval for 5 v | ience interval for 5 v | aence interval for 5 v | dence interval for 5 v | idence interval for 5 v | idence interval for 5 v | ndence interval for Sv | fidence interval for 5 v | maence interval for 5 v | ifidence interval for 5 v | nfidence interval for Sv | nfidence interval for 5 v | ntidence interval for 5 v |
| ı | ı | r | K | KI | KI | KI | KI | KI | KI | KI | KI | KI | K | K | K | K | K | K | K | K | K | K | K | K | K | K | K | K | K | K | ı | ľ | 1 | 4 | | | | | į | | ١ | ١ | ١ | ١ | ١ | ١, | ١( | ١( | ۱ د | ١د | ٥١ | ٥ د | ٥ ( | ٥ ر | ٥, | ٥١ | ٥١ | ٥, | 21 | 21 | 21 | 21 | 21 | · 51 | · 51 | rδı | r 51 | )r 51 | or 51 | or 51 | or 51 | or 51 | or 51 | or 51 | ror 5 v | tor 5 v | tor 21 | tor 21 | tor 21 | 101 21 | 101 21 | 1 tor 21 | II TOR 51 | ai tor 5 v | ai tor Sv | ai for 5 v | al for 5 | ai for 51 | vai for 5 v | vai for 5 v | rvai for 5 v | rvai for 5 v | rval for 5 v | ervai for 5 v | erval for 5 v | ervai for 5 v | terval for 5 v | tervai for 5 v | itervai for 5 v | itervai for 5 v | nterval for 5 v | intervai for 5 v | interval for 51 | interval for 5 v | e interval for 51 | e interval for 51 | e interval for 51 | ce interval for 51 | ce interval for 51 | ice interval for 51 | ice interval for 5 v | nce interval for 5 v | ince interval for 51 | ence interval for 51 | ence interval for 51 | ence interval for 51 | ience interval for 5 v | aence interval for 51 | dence interval for 51 | idence interval for 51 | idence interval for 51 | ridence interval for 51 | fidence interval for 51 | maence interval for 51 | ifidence interval for 51 | ntidence interval for 5 v | nfidence interval for 51 | ntidence interval for 51 |

| Number of | SVR12 rates | 95% | 6 Confidence Ir | nterval* |
|-----------|-------------|-------------|--------------------|----------|
| patients | | Lower Limit | <b>Upper Limit</b> | Width |
| 200 | 90% | 85.1 | 93.4 | 8.4% |
| 200 | 95% | 91.0 | 97.3 | 6.2% |
| 225 | 90% | 85.4 | 93.3 | 7.9% |
| 225 | 95% | 91.3 | 97.2 | 5.8% |
| 235 | 90% | 85.6 | 93.2 | 7.7% |
| 235 | 95% | 91.4 | 97.1 | 5.7% |

<sup>\*</sup> two-sided 95% confidence interval according the Wilson Score method

### 9.6 Data Management

### 9.6.1 Electronic Case Report Forms

Data for this study will be recorded in English by each participating center via an electronic data capture (EDC) system using a web-based eCRF. Examinations, diagnostic measures, laboratory assessments, findings and observations routinely performed in patients with CHC included in this cohort, will be transcribed by the investigator or designee from the source documents into the eCRF. Only data specified in the protocol will be entered into the eCRF. For each enrolled patient, the investigator or designee will create a new patient file in the eCRF and a unique patient number will be automatically allocated by the system.

A comprehensive data validation program utilizing front-end checks in the eCRF will validate the data. Automated checks for data consistency will be implemented, discrepancies need to be solved by the researcher in the eCRF before the module can be completed.

Follow-up on eCRF data for medical plausibility will be done by AbbVie personnel (or their representatives). Queries will be generated in the eCRF for online resolution at the site. The investigator or an authorized member of the investigator's staff will make any necessary data corrections to the eCRF. All change information, including the date and person performing the corrections, will be available via the audit trail, which is part of the EDC system. The principal investigator of each site will finally review the eCRFs for completeness and accuracy of available data and provide his or her electronic signature and date to the eCRFs as evidence thereof.

Access to the EDC system will be provided for the duration of the study through a password-protected method of internet access. Such access will be removed from investigator sites at the end of the site's participation in the study. Data from the EDC system will be archived on appropriate data media (e.g. CD-ROM) and provided to the investigator as a durable record of the site's eCRF data.

Original Questionnaires will be sent from the participating site to:

| Name: |
|----------|
| Address: |
| Tel.: |
| Fax: |

### 9.6.2 Assignment of Preferred Terms

AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and will be tabulated by primary MedDRA system organ class (SOC) and preferred term (PT). For treatments, surgical and medical procedures the international non-proprietary name (INN) Drug Terms and Procedures Dictionary will be used.

### 9.7 Data Analysis

# 9.7.1 Analysis Population, Time Windows and Handling of Missing Data

The target population (TP) is defined as all patients who fulfill the criteria specified in Section 9.2.1. The core population (CP) is defined as all patients of the TP, who have started the treatment combination recommended in the current local label for their disease characteristics. Patients not receiving the treatment recommended in the local label will be summarized in the non-core population (NCP). In addition, the core population with sufficient follow-up data (CPSFU) is defined as all CP patients, who fulfil one of the following criteria:

- (1) evaluable HCV RNA data ≥70 days after the last actual dose of the ABBVIE REGIMEN (i.e. data within the SVR12 time window)
- (2) a HCV RNA value ≥50 IU/mL at the last measurement post-baseline (i.e. no virological response achieved at the last measurement on-treatment or posttreatment)
- (3) HCV RNA <50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥70 days after the last actual dose of the ABBVIE REGIMEN due to reasons related to safety (e.g. dropped out due to AE) or incomplete efficacy information (e.g. virologic failure such as relapse is reported in the eCRF but date and value of the corresponding HCV RNA test is missing). This means only patients who had virological response at their last on-treatment or post-treatment measurement, but had no HCV RNA measurements ≥70 days post-treatment for reasons not related to safety or effectiveness (e.g. lost-to-follow-up or patient not willing to perform an additional HCV RNA test ≥70 days post-treatment) will be excluded from this analysis.

The Safety Population (SP) is defined as all patients who received at least one dose of the ABBVIE REGIMEN.

In accordance with the non-interventional nature of the study all HCV RNA measurements will be performed at the sole discretion of the physician and all HCV RNA measurements have to be entered into the eCRF. All recorded HCV RNA values will be assigned to appropriate time points (baseline, on-treatment visits, EoT visit, post-treatment visits). The time windows for the assignments will be specified in the statistical analysis plan (SAP).

No data will be imputed for any effectiveness or safety analyses except for the analyses of the HCV RNA endpoints. When there is no HCV RNA value in a visit time window post-baseline, but prior to EoT, the closest values before and after the window, regardless of the value chosen for the subsequent and preceding window, will be used for the flanking imputation described below. If a patient has a missing HCV RNA value at a post-baseline visit prior to EoT but has undetectable HCV RNA (with LLoD ≤50 IU/mL) or unquantifiable, but detectable HCV RNA levels (with LLoQ ≤50 IU/mL) at both the preceding and succeeding measurements, the HCV RNA level will be considered undetectable or unquantifiable, respectively, at this visit for this patient. In addition, if a patient has an unquantifiable HCV RNA level at the preceding measurement and an undetectable HCV RNA level at the succeeding measurement, or vice versa, the HCV RNA level will be imputed as unquantifiable at this visit for this patient. For virological response at EoT a corresponding backward imputation approach will be applied. This means if HCV RNA is missing at EoT, then unquantifiable or undetectable will be assumed for EoT, if the succeeding HCV RNA value is undetectable or unquantifiable. For SVR12 the single last available HCV RNA measurement within 70 -126 days posttreatment will be used. For SVR analysis, if there is no value in this time window, but there is an HCV RNA value after the window, then it will be imputed into the SVR window. Subsequent to this flanking and backward imputation, if the HCV RNA value remains missing at a specific time point, then the patients will considered as virological failure at this time point (i.e. not undetectable or unquantifiable).

### 9.7.2 Demographics and Disease Characteristics

All baseline and disease characteristics will be summarized for the CP stratified by the CP analysis groups (i.e. based on genotype and fibrosis status), which are relevant for scheduled treatment combination (ABBVIE REGIMEN ± RBV). In addition, baseline summaries will be repeated for the SP and the TP. Summary statistics (n, mean, median, standard deviation [SD], and range) will be generated for continuous variables (e.g. age and body mass index [BMI]). The number and percentage of patients will be presented for categorical variables (e.g. gender and race). Further details of analysis populations and the CP analysis groups will be specified in the SAP, taking into account the ABBVIE REGIMEN recommended in the current local label for various patient groups.

### 9.7.3 Effectiveness Analysis

The primary effectiveness analysis on clinical outcomes will be performed on all patients in the CP stratified by the CP analysis groups. Due to the non-interventional nature of this study several different methods for determination of the HCV RNA value can be applied. For the purpose of the statistical analysis, a HCV RNA measurement is considered ≤50 IU/mL.

- if a PCR test was used
- and the test result is undetectable and the LLoD of the test is ≤50 IU/mL or the test result is unquantifiable and the LLoQ is ≤50 IU/mL

### 9.7.3.1 Primary Effectiveness Endpoint

The percentage of patients achieving SVR12 (HCV RNA <50 IU/mL 12 weeks [i.e. at least 70 days] after the last actual dose of the ABBVIE REGIMEN) is the primary effectiveness endpoint.

### 9.7.3.2 Secondary Effectiveness Endpoints

The secondary effectiveness endpoints are:

- The percentage of patients with virological response (HCV RNA <50 IU/mL) at EoT
- The percentage of patients with relapse (defined as HCV RNA <50 IU/mL at EoT followed by HCV RNA ≥50 IU/mL)
- The percentage of patients with breakthrough (defined as at least one documented HCV RNA <50 IU/mL followed by HCV RNA ≥50 IU/mL during treatment).
- The number and percentage of patients meeting each and any of the following SVR12 non-response categories:
  - On-treatment virologic failure (breakthrough [defined as above ] or failure to suppress [each measured on-treatment HCV RNA value ≥50 IU/mL])
  - Relapse (defined as HCV RNA <50 IU/mL at EoT or at the last ontreatment HCV RNA measurement followed by HCV RNA ≥50 IU/mL post-treatment)

- Premature study drug discontinuation with no on-treatment virologic failure
- Missing SVR12 data and/or none of the above criteria

### 9.7.3.3 Statistical Methods for Analysis of Effectiveness Variables

The simple percentage of patients achieving SVR12 will be calculated and a two-sided 95% confidence interval (CI) of the percentage will be computed based on the Wilson score method.

Corresponding methods will be used for other response rates (EoT response rate, relapse rate, viral breakthrough). The relapse rates will be estimated in patients of the CP analysis groups with EoT response and sufficient HCV RNA measurements post-treatment. Viral breakthrough rates will be estimated in all patients of the CP analysis groups, who have at least one undetectable HCV RNA measurement on-treatment and at least one on-treatment or EoT measurement thereafter.

Univariate and multiple logistic regression (MLR) methods will be used to investigate the impact of the following explanatory covariates on SVR12:

- Key demographic information
- Mode of CHC infection
- HCV RNA level at baseline
- Most recent stage of liver fibrosis
- HCV genotype and subtype (if available)
- Type of treating institute
- Liver and/or CHC related co-morbidities
- Key clinical chemistry and hematology laboratory variables at baseline
- In treatment experienced patients only:
  - Most recent prior treatment for CHC
  - Outcome of most recent prior CHC treatment

Further details and additional covariates will be specified in the SAP.

These analyses will be of exploratory nature, data driven, and will be repeatedly performed for various CP Analysis Groups, since not each covariate might be predictive in each patient group. Furthermore, the fact that treatment regimens will differ in the various patient groups has to be taken into account, when selecting the patient groups for each MLR analysis. Backward selection procedures will be applied to generate the final MLR models and a p-value <0.05 will be used for the covariates to stay in the model in a

backward elimination step. Logistic regression methods will also be used to investigate the impact of treatment adherence on SVR12.

### 9.7.4 Clinical Laboratory Data

All reported clinical laboratory test results will be assigned to one of the time points using the time windows specified in the table below.

**Table 4 - Analysis Time Windows** 

| Phase | Time point | Time Window |
|---|---|---|
| Pre-Treatment | Baseline | Last value prior to start of study treatment |
| | | (i.e. ≤study day 1) |
| | | Study day during treatment period |
| | | (Study day 1 = first treatment day) |
| Treatment Weeks | 4 (day 29) | 15 - 42 |
| | 8 (day 57) | 43 - 70 |
| | 12 (day 85) | 71 - 98 |
| | 16 (day 113) | 99 - 126 |
| EoT | Actual EoT | Study day of last dose |
| | | (28 days prior to EoT - 14 days post EoT) |
| Post Treatment | 4 weeks | 15 – 56 post EoT |
| | (day 29 post EoT) | |
| | 12 weeks | 57 – 126 post EoT |
| | (day 85 post EoT) | |
| | 24 weeks | 127 – 252 post EoT |
| | (day 169 post EoT) | |

Mean changes from baseline to each post-baseline visit will be summarized descriptively.

Laboratory data values collected during the treatment period will be categorized as low, normal, or high based on reference ranges used in this study. The number and percent of patients who experience post-baseline shifts during treatment in clinical laboratory values from low/normal to high and high/normal to low based on the reference range will be summarized.

Additional details of the analyses of clinical laboratory data will be specified in the SAP.
#### 9.7.5 PSP and PAM

The contribution of the patient support program (PSP) to disease control, treatment continuation over time, patient satisfaction and PSP utilization will be analyzed using descriptive and exploratory statistical methods. Appropriate frequency tables will summarize all corresponding variables of the PSP questionnaires (see ANNEX 2 and 3) over time stratified by ABBVIE REGIMEN arms. In addition, multiple logistic regression (MLR) analysis will be performed to investigate the association between the use of the PSP, the patient satisfaction variables of the PSP questionnaires with the probability to treatment completion. These MLRs will be performed similar to the MLRs for SVR12 (see Section ). Additional details will be specified in the SAP.

The Patient Activation Measure (PAM) 13 item scale is a measure used to assess the patient knowledge, skill, and confidence for self-management. Each of the 13 items can be answered with one of four possible response options, which are "disagree strongly" (1), "disagree" (2), "agree" (3), "agree strongly" (4).

Based on responses to the 13-item measure, the score is calculated by adding up the raw scores (range of the sum: 13 - 52) and mapping up the value onto a scale of 0–100 indicating strength of agreement with the 13 items (100 \* (sum - 13) / (52 - 13)). The final score can be assigned to one of the four levels of activation. A higher score indicates that the patient is likely to participate more actively in health care processes and takes more responsibility for his or her health.

In case of missing item values, the mean value of the available items will be used for replacement. However, if there are less than nine items answered, no summary score will be calculated.

A summary table will show descriptive statistics (n, mean, median, SD, minimum and maximum) of the score for baseline and EoT, as well as change from baseline. In addition analysis of covariance (ANCOVA) will be applied to investigate the effect of the different ABBVIE REGIMENS (± RBV) on the activation score using the corresponding score at baseline as covariate. Further details will be specified in the SAP.

#### 9.7.6 Tolerability Analysis

All tolerability variables will be summarized using descriptive statistical methods for the SP stratified by type of combination treatment.

All SAEs, non-serious AEs and pregnancy occurrences are to be reported for patients included in the study (see Section 11.0 and 9.2.3). AEs will be coded using MedDRA.

The number and percentage of patients with treatment-emergent AEs (i.e. any reported event that begins or worsens in severity after initiation of study drug through 30 days post-study drug dosing) will be tabulated by primary MedDRA SOC and PT. Corresponding summary tables will be provided for all serious treatment-emergent AEs. The tabulation of the number of patients with treatment-emergent AEs by severity and relationship to study drug will also be provided. Patients reporting more than one AE for a given MedDRA PT will be counted only once for that term using the most severe incident for the severity summary table and the most related for the relationship summary table. Patients reporting more than one type of event within a SOC will be counted only once for that SOC.

Additional details of the analysis of AEs will be specified in the SAP.

#### 9.7.7 Interim Assessments

No interim assessments are planned.

#### 9.8 Quality Control

The sites will be instructed in the protocol, the functionality and handling of the eCRF, and the requirement to maintain source documents for each patient in the study (see Section 9.4).

A comprehensive data validation program utilizing front-end checks in the eCRF will validate the data. Automated checks for data consistency will be implemented, discrepancies need to be solved by the researcher in the eCRF before the module can be completed. Follow-up on eCRF data for medical plausibility will be done by AbbVie personnel (or their representatives). The principal investigator of each site will finally review the eCRFs for completeness and accuracy of available data and provide his or her electronic signature and date to eCRFs as evidence thereof.

Continuous monitoring of the study and frequent site telephone contacts will be done by AbbVie or a CRO working on behalf of AbbVie.

#### 9.9 Limitations of the Research Methods

The limitations of observational studies, such as uncontrolled confounding by lack of randomization, and difficulties to clearly interpret treatment effects in the context of missing data are well known. Their validity can be increased by accurate outcome measurements, documentation of the most common confounders, sufficient length of follow-up and by activities to obtain complete recording of available data as well as by searches for missing key data.

The most important outcome measure in this study is HCV RNA. Missing or unrecorded follow-up HCV RNA data can in particular lead to an underestimation of the real SVR rate as compared to the SVR rate of interventional trials. Highly sensitive and quantitative diagnostic tests are required to measure HCV RNA levels in blood. In an observational study each center will be using its own test – either commercially available or so-called "home-brew" tests – which might change from one visit to the next within a patient data set. The challenge is to accurately and consistently document test properties such as the LLoD and the LLoQ to put the results into perspective of prior outcomes from randomized controlled trials with (usually) central laboratory assessments for all trial participants.

#### 10.0 Protection of Human Subjects

This observational study will be run in compliance with local laws and regulations. Notification/submission to the responsible regulatory authorities, Ethics Committee (EC) and/or Competent Authorities (CAs) will be done as required by local laws and regulations.

The investigator is responsible to ensure that written patient informed consent will be obtained prior to patient inclusion

To maintain patient confidentiality, no demographic data that can identify the patient will be collected (e.g. initials, date of birth) - only the patient age will be collected. In order to protect patient identity, a unique number will be assigned to each patient and related study recording.

#### 11.0 Management and Reporting of Complaints

A Complaint is any written, electronic, or oral communication that alleges deficiencies related to the physical characteristics, identity, quality, purity, potency, durability, reliability, safety, effectiveness, or performance of a product/device after it is released for distribution.

Complaints associated with any component of the ABBVIE REGIMEN must be reported to the Sponsor (11.2.2).

For adverse events, please refer to Sections 11.1.1 through 11.1.6. For product complaints, please refer to Section 11.2.

#### 11.1 Medical Complaints

PRO data are not considered a potential source of adverse reactions. However, participating sites should review the PRO data and if a possible product-related event (including a suspected adverse reaction) is noted, the HCP must determine whether the event is related to the ABBVIE REGIMEN ± RBV (or any other AbbVie authorized product) and if so, it should be reported to AbbVie.

Medication errors (this refers to any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in control of the HCP, patient or consumer) should be reported by the HCP to AbbVie.

The relevant AbbVie Pharmacovigilance contact details are specified below:

| Name: |
|----------|
| Address: |
| Tel.: |
| Fax: |
| Email: |

### 11.1.1 Adverse Event Definition and Serious Adverse Event Categories

An adverse event (AE) is defined as any untoward medical occurrence in a patient, which does not necessarily have a causal relationship with their treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not the event is considered causally related to the use of the product.

Such an event can result from use of the drug as stipulated in the labeling, as well as from accidental or intentional overdose, drug abuse, or drug withdrawal. Any worsening of a pre-existing condition or illness is considered an AE.

If an AE meets any of the following criteria, it is considered a serious adverse event (SAE):

**Death of Patient:** An event that results in the death of a patient.

Life-Threatening: An event that, in the opinion of the investigator, would

> have resulted in immediate fatality if medical intervention had not been taken. This does not include an event that would have been fatal if it had

occurred in a more severe form.

**Hospitalization:** An event that results in an admission to the hospital

> for any length of time. This does not include an emergency room visit or admission to an outpatient

facility.

**Prolongation of** An event that occurs while the study patient is Hospitalization:

hospitalized and prolongs the patient's hospital stay.

**Congenital Anomaly:** An anomaly detected at or after birth, or any anomaly

that results in fetal loss.

**Persistent or Significant** 

Disability/Incapacity:

An event that results in a condition that substantially interferes with the activities of daily living of a study

patient. Disability is not intended to include

experiences of relatively minor medical significance such as headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g. sprained

ankle).

**Important Medical Event** Requiring Medical or Surgical Intervention to **Prevent Serious Outcome:** 

An important medical event that may not be immediately life-threatening or result in death or hospitalization, but based on medical judgment may jeopardize the patient and may require medical or surgical intervention to prevent any of the outcomes listed above (i.e. death of patient, life threatening, hospitalization, prolongation of hospitalization, congenital anomaly, or persistent or significant disability/incapacity). Additionally, any elective or

spontaneous abortion or stillbirth is considered an important medical event. Examples of such events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

#### 11.1.2 Severity

The following definitions will be used to rate the severity for any AE being collected as an endpoint/data point in the study and for all SAEs.

**Mild:** The AE is transient and easily tolerated by the patient.

**Moderate:** The AE causes the patient discomfort and interrupts the patient's

usual activities.

**Severe:** The AE causes considerable interference with the patient's usual

activities and may be incapacitating or life threatening.

#### 11.1.3 Relationship to Pharmaceutical Product

The following definitions will be used to assess the relationship of the AE to the use of product:

**Reasonable Possibility** An AE where there is evidence to suggest a causal

relationship between the product and the AE.

**No Reasonable** An AE where there is no evidence to suggest a causal

**Possibility** relationship between the product and the AE.

If no reasonable possibility of being related to product is given, an alternate etiology must be provided for the AE.

#### 11.1.4 Serious Adverse Event Collection Period

SAEs will be reported to AbbVie from the time the physician obtains the patient's informed consent until 30 days or 5 half-lives following the intake of the last dose of physician-prescribed treatment.

#### 11.1.5 Serious and non-serious Adverse Event Reporting

In the event of an **SAE**, the physician will:

- For events from patients using the ABBVIE REGIMEN ± RBV (or any other AbbVie authorized product) report to AbbVie within 24 hours of the physician becoming aware of the event by using the eCRF system or notifying the AbbVie contact person identified in Section 11.0.
- For events from patients using a non-AbbVie product notify the Marketing Authorization Holder (MAH) of the product within 24 hours of the physician becoming aware of the event.

In the event of a *non-serious AE*, the physician will:

 For events from patients using the ABBVIE REGIMEN ± RBV report to AbbVie by using the eCRF system.

#### 11.1.6 Pregnancy Reporting

Patients and their partners should avoid pregnancy and males should avoid sperm donation throughout the course of the HCV treatment and for 30 days after the end of treatment with DAAs only, or for 7 months after the last dose of RBV (or per local RBV label) and/or consistent with local treatment guidelines for RBV.

In the event of a pregnancy occurrence in the patient, the physician will report to AbbVie within 24 hours of the physician becoming aware of the pregnancy by using the eCRF system or notifying the AbbVie contact person identified in Section 11.0.

The investigator is encouraged to report the pregnancy information to the voluntary RBV Pregnancy Registry, if RBV is included within the regimen.

#### 11.2 Product Complaint

#### 11.2.1 Definition

A Product Complaint is any Complaint (see Section **** for the definition) related to the drug or drug component of the product.

For a product this may include, but is not limited to, damaged/broken product or packaging, product appearance whose color/markings do not match the labeling, labeling discrepancies/inadequacies in the labeling/instructions (example: printing illegible), missing components/product, or packaging issues.

#### 11.2.2 Reporting

The relevant AbbVie Product Complaint contact details are specified below:

| Name: |
|----------|
| Address: |
| Tel.: |
| Fax: |
| Email: |

Product Complaints concerning the ABBVIE REGIMEN must be reported to the Sponsor within 24 hours of the study site's knowledge of the event via local Product Complaint reporting practices. Product Complaints occurring during the study will be followed-up to a satisfactory conclusion. All follow-up information is to be reported to the Sponsor (or an authorized representative) and documented in source as required by the Sponsor. Product Complaints associated with adverse events will be reported in the study summary. All other complaints will be monitored on an ongoing basis.

Product complaints involving a non-Sponsor investigational product and/or device should be reported to the identified contact or manufacturer, as necessary per local regulations.

Product Complaints may require return of the product with the alleged complaint condition. In instances where a return is requested, every effort should be made by the investigator to return the product within 30 days. If returns cannot be accommodated within 30 days, the site will need to provide justification and an estimated date of return.

The description of the complaint is important for AbbVie in order to enable AbbVie to investigate and determine if any corrective actions are required.

### 12.0 Plans for Disseminating and Communicating Study Results

At the end of this observational study, a report will be written by AbbVie or a CRO working on behalf of AbbVie. The required standard study report template will be followed. This report will contain a description of the objectives of the study, the methodology and its results and conclusions. The completed eCRFs, [patient questionnaires, interim assessments], the final study output and study report are the confidential property of AbbVie and may not be released to unauthorized people in any form (publications or presentations) without express written approval from AbbVie. The study results will be submitted to local authorities by the participating countries per local laws and regulations.

The results of this study will be made publicly available on one of the primary registries in the World Health Organization (WHO) Registry Network which meet the requirements of the ICMJE (International Committee of Medical Journal Editors) and through scientific publications. Authorship will be in line with ICMJE' authorship requirements [68].

#### 13.0 References

- [1] Lozano R, Naghavi M, Foreman K, et al. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet 2012; 380: 2095-128.
- [2] Chen SL, Morgan TR. The natural history of hepatitis C virus (HCV) Infection. Int J Med Sci 2006; 3: 47-52.
- [3] Hoofnagle JH. Course and outcome of hepatitis C. Hepatology 2002; 36 (Suppl 1): S21-9.
- [4] Di Bisceglie AM. Natural history of hepatitis C: its impact on clinical management. Hepatology 2000; 31: 1014-8.
- [5] Pawlotsky JM. Hepatitis C virus: from discovery to eradication in 40 years? Clin Microbiol Infect 2011; 17: 105-6.
- [6] Lavanchy D. Evolving epidemiology of hepatitis C virus. Clin Microbiol Infect 2011; 17: 107-15.
- [7] WHO. Weekly epidemiological record. 2000; 75, 17-28. Available at http://www.who.int/docstore/wer/pdf/2000/wer7503.pdf.
- [8] Szabo SM, Bibby M, Yuan Y et al. The epidemiologic burden of hepatitis C virus infection in Latin America. Ann Hepatol 2012; 11: 623-35.
- [9] Pereira LMMB, Martelli CMT, Moreira RC et al. Prevalence and risk factors of hepatitis C virus infection in Brazil, 2005 through 2009: a cross-sectional study. BMC Infect Dis 2013; 13: 1-12.
- [10] Eurosurveillance 2003; 8 (5): 99-118.
- [11] Smith DB, Bukh J, Kuiken C, et al. Expanded classification of hepatitis C virus into 7 genotypes and 67 subtypes: updated criteria and genotype assignment web resource. Hepatology 2014; 59: 318-27.
- [12] US Department of Health and Human Services Centers for Disease Control and Prevention. Recommendations for prevention and control of hepatitis C virus (HCV) infection and HCV related chronic disease. CDC Report1998; 47: 1-39
- [13] Houghton M. Hepatitis C viruses. In: Fields BN, Knipe DM, Howley PM, eds, Fields Virology (3rd ed). Philadelphia: Lippincott Raven, 1996: 1035-58.
- [14] Global surveillance and control of hepatitis C. Report of a WHO Consultation organized in collaboration with the Viral Hepatitis Prevention Board, Antwerp, Belgium. J Viral Hepat 1999; 6: 35-47.
- [15] WHO. HCV genotypes. Available at http://www.who.int/csr/disease/hepatitis/whocdscsrlyo2003/en/index2.html#genome; accessed July 07, 2014.
- [16] Prati D. Transmission of hepatitis C virus by blood transfusions and other medical procedures: a global review. J Hepatol 2006; 45: 607-16.

- [17] Central and Eastern European Harm Reduction Network (CEEHRN). Hepatitis C among drug users in the new EU member states and neighborhood:

  Recommendations for action. CEEHRN brochure/leaflet 2006. Available at http://www.aidsactioneurope.org/clearinghouse/topics/hepatitis-c-among-drug-users-new-eu-member-states-and.
- [18] Alberti A, Chemello L, Benvegnù L. Natural history of hepatitis C. J Hepatol 1999; 31 (Suppl 1): 17-24.
- [19] Alazawi W, Cunningham M, Dearden J, Foster GR. Systematic review: outcome of compensated cirrhosis due to chronic hepatitis C infection. Aliment Pharmacol Ther 2010; 32: 344-55.
- [20] Brown RS. Hepatitis C and liver transplantation. Nature 2005; 436: 973-78.
- [21] Villano SA, Vlahov D, Nelson KE, Cohn S, Thomas DL. Persistenc of viremia and the importance of long-term follow-up after acute hepatitis C infection. Hepatology 1999; 29: 908-14.
- [22] Thomas DL, Astemborski J, Rai RM, et al. The natural history of hepatitis C virus infection: host, viral, and environmental factors. JAMA 2000; 284: 450-6.
- [23] Dore GJ, Ward J, Thursz M. Hepatitis C disease burden and strategies to manage the burden (Guest Editors Mark Thursz, Gregory Dore and John Ward). J Viral Hepat 2014; 21 (Suppl 1): 1-4.
- [24] Davis GL, Albright JE, Cook SF, Rosenberg DM. Projecting future complications of chronic hepatitis C in the United States. Liver Transpl 2003; 9: 331-8.
- [25] Strader DB, Wright T, Thomas DL, Seeff LB. AASLD practice guidelines: diagnosis, management, and treatment of hepatitis C. Hepatology 2004; 39: 1147-70.
- [26] Dienstag LJ, McHutchison JG. American gastroenterological association technical review on the management of hepatitis C. Gastroenterology 2006; 130: 231-64.
- [27] Ghany MG, Strader DB, Thomas DL, Seeff LB. AASLD practice guidelines: diagnosis, management, and treatment of hepatitis C: an update. Hepatology 2009; 49: 1335-74.
- [28] Backus LI, Boothroyd DB, Phillips BR, et al. A sustained virologic response reduces risk of all-cause mortality in patients with hepatitis C. Clin Gastroenterol Hepatol 2011; 9: 509-16.
- [29] Van der Meer AJ, Veldt BJ, Feld JJ, et al. Association between sustained virological response and all-cause mortality among patients with chronic hepatitis C and advanced hepatic fibrosis. JAMA 2012; 308: 2584-93.
- [30] Everson GT, Balart L, Lee SS, et al. Histological benefits of virological response to peginterferon alfa-2a monotherapy in patients with hepatitis C and advanced fibrosis or compensated cirrhosis. Aliment Pharmacol Ther 2008; 27: 542-51.
- [31] Poynard T, McHutchison JG, Manns M, et al. Impact of pegylated interferon alfa-2b and ribavirin on liver fibrosis in patients with chronic hepatitis C. Gastroenterology 2002; 122: 1303-13.
- [32] Shiffman M, Hofmann CM, Thompson EB, et al. Relationship between biochemical, virologic and histologic response during interferon treatment of chronic hepatitis C. Hepatology 1997; 26: 780-5.

- [33] Bruno S, Stroffolini T, Colombo M, et al. Sustained virological response to interferonalpha is associated with improved outcome in HCV-related cirrhosis: a retrospective study. Hepatology 2007; 45: 579-87.
- [34] Di Bisceglie AM, Shiffman M, Everson GT, et al. Prolonged antiviral therapy with peginterferon to prevent complications of advanced liver disease associated with hepatitis C: results of the hepatitis C antiviral long-term treatment against cirrhosis (HALT-C) trial. Hepatology 2007; 46 (Suppl S1): 290A.
- [35] Camma C, Di Bona D, Schepis F, et al. Effect of peginterferon alfa-2a on liver histology in chronic hepatitis C: a meta-analysis of individual patient data. Hepatology 2004; 39: 333-42.
- [36] McHutchison JG, Gordon SC, Schiff ER, et al. Interferon alfa-2b alone or in combination with ribavirin as initial treatment for chronic hepatitis C. Hepatitis Interventional Therapy Group. NEJM 1998; 339: 1485-92.
- [37] Zeuzem S, Feinman SV, Rasenack J, et al. Peginterferon α-2a in patients with chronic hepatitis C. NEJM 2000; 343: 1666-72.
- [38] Poynard T, McHutchison JG, Goodman Z, Ling MH, Albrecht J. Is an "à la carte" combination interferon alfa-2b plus ribavirin regimen possible for the first line treatment in patients with chronic hepatitis C? Hepatology 2000; 31: 211-8.
- [39] Fried MW, Shiffman M, Reddy KR, et al (for the PEGASYS<sup>®</sup> International Study Group). Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. NEJM 2002; 347: 975-82.
- [40] Manns M, McHutchison JG, Gordon SC et al. PegInterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomized trial. Lancet 2001; 358: 958-65.
- [41] Hadziyannis SJ, Sette H Jr, Morgan TR et al. Peginterferon-alpha 2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med 2004: 140: 346-55.
- [42] Jacobson IM, McHutchison JG, Dusheiko GM et al. Telaprevir in combination with peginterferon and ribavirin in genotype 1 HCV treatment-naive patients: final results of phase 3 ADVANCE study. Hepatology 2010; 52 (Suppl S1): 427A.
- [43] Sherman KE, Flamm SL, Afdhal NH et al. Telaprevir in combination with peginterferon alfa2b and ribavirin for 24 or 48 weeks in treatment-naive genotype 1 HCV patients who achieved an extended rapid viral response: final results of Phase 3 ILLUMINATE study. Hepatology 2010; 52 (Suppl S1): 401A.
- [44] Poordad F, McCone J, Bacon BR et al. Boceprevir (BOC) combined with peginterferon alfa-2b/ribavirin (P/R) for treatment-naive patients with hepatitis C (HCV) genotype 1: SPRINT-2 final results. Hepatology 2010; 52 (Suppl S1): 402A.
- [45] EASL Recommendations on Treatment of Hepatitis C 2014. J Hepatol 2014; doi: 10.1016/j.jhep.2014.05.001 (Epub ahead of print).
- [46] AASLD. Recommendations for Testing, Managing, and Treating Hepatitis C. 2014: 1-50. Available at http://www.hcvguidelines.org/sites/default/files/full\_report.pdf.

- [47] Jacobson IM, Dore G, Foster G et al. Simeprevir with pegylated interferon alfa 2a plus ribavirin in treatment-naive patients with chronic hepatitis C virus genotype 1 infection (QUEST-1): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet 2014; doi: 10.1016/S0140-6736(14)60494-3 (Epub ahead of print).
- [48] Manns M, Marcellin P, Poordad F, et al. Simeprevir with pegylated interferon alfa 2a or 2b plus ribavirin in treatment-naive patients with chronic hepatitis C virus genotype 1 infection (QUEST-2): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet 2014; doi: 10.1016/S0140-6736(14)60538-9 (Epub ahead of print).
- [49] Forns X, Lawitz E, Zeuzem S, et al. Simeprevir with Peginterferon and ribavirin leads to high rates of SVR in patients with HCV genotype 1 who relapsed after previous therapy: a phase 3 trial. Gastroenterology. 2014; 146: 1669-79.
- [50] Reddy KR, Zeuzem S, Zoulim F, et al. A Phase III randomised, double-blind study to evaluate the efficacy, safety and tolerability of simeprevir vs telaprevir in combination with pegylated interferon and ribavirin in chronic hepatitis C virus genotype 1 treatment-experienced patients: the ATTAIN study. Abstract APASL 2014 Brisbane, Australia. Available at http://www.natap.org/2014/APASL/APASL 20.htm.
- [51] Full prescribing information Olysio. Available at http://www.olysio.com/shared/product/olysio/prescribing-information.pdf; accessed February 09, 2014.
- [52] Lawitz E, Mangia A, Wyles D, et al. Sofosbuvir for previously untreated chronic hepatitis C infection. NEJM 2013; 368: 1878-87.
- [53] Lalezari L, Nelson D, Hyland R, et al. Once daily sofosbuvir plus ribavirin for 12 and 24 weeks in treatment-naive patients with HCV infection: the QUANTUM study. J Hepatol 2013; 58 (Suppl 1): S346.
- [54] Osinusi A, Meissner EG, Lee YJ, et al. Sofosbuvir and ribavirin for hepatitis C genotype 1 in patients with unfavorable treatment characteristics: a randomized clinical trial. JAMA 2013; 310: 804-11.
- [55] Menon RM, Klein CE, Lawal AA, et al. Pharmacokinetics and tolerability of the HCV protease inhibitor ABT-450 following single ascending doses in healthy adult volunteers with and without ritonavir. Abstract of HepDART 2009, Kohala Coast, Hawaii, USA. Available at http://www.natap.org/2009/hepDART/hepDART\_03.htm.
- [56] Feld JJ, Kowdley KV, Coakley E, et al. Treatment of HCV with ABT-450/r ombitasvir and dasabuvir with ribavirin. NEJM 2014; 370: 1594-603.
- [57] Zeuzem S, Jacobson IM, Baykal T, et al. Retreatment of HCV with ABT-450/r-ombitasvir and dasabuvir with ribavirin. NEJM 2014: 370: 1604-14.
- [58] Andreone P, Colombo MG, Enejosa JV, et al. ABT-450, ritonavir, ombitasvir, and dasabuvir achieves 97% and 100% sustained virologic response with or without ribavirin in treatment-experienced patients with HCV genotype 1b infection. Gastroenterology 2014; doi: 10.1053/j.gastro.2014.04.045 (Epub ahead of print).
- [59] Ferenci P, Bernstein D, Lalezari J, et al. ABT-450/r-ombitasvir and dasabuvir with or without ribavirin for HCV. NEJM 2014; 370: 1983-92.
- [60] Poordad F, Hezode C, Trinh R, et al. ABT-450/r-ombitasvir and dasabuvir with ribavirin for hepatitis C with cirrhosis. NEJM 2014; 370: 1973-82.

- [61] Hezode C, Marcellin P, Pol S, et al. Results from the phase 2 PEARL-I study: interferon-free regimens of ABT-450/R + ABT-267 with or without ribavirin in patients with HCV genotype 4 infection. J Hepatol 2014; 60 (Suppl 1): S24.
- [62] Hezode C, Fontaine H, Dorival C et al. Effectiveness of telaprevir or boceprevir in treatment-experienced patients with HCV genotype 1 infection and cirrhosis. Gastroenterology 2014; 147: 132-42.
- [63] Colombo M, Fernández I, Abdurakhmanov D, et al. Safety and on-treatment efficacy of telaprevir: the early access programme for patients with advanced hepatitis C. Gut 2014; 63: 1150-8.
- [64] Marley J. Efficacy, effectiveness, efficiency. Aust Prescr 2000; 23: 114-5.
- [65] Singal AG, Higgins PDR, Waljee AK. A primer on effectiveness and efficacy trials. Clin Trans Gastroenterol 2014; 5 (e45): 1-4.
- [66] Marcellin P, Cheinquer H, Curescu M, et al. High sustained virologic response rates in rapid virologic response patients in the large real-world PROPHESYS cohort confirm results from randomized clinical trials. Hepatology 2012; 56: 2039-50.
- [67] Thompson AJ, Muir AJ, Sulkowski MS, et al. IL28B polymorphism improves viral kinetics and is the strongest pre-treatment predictor of SVR in HCV-1 patients. Gastroenterology 2010; 139: 120-9.
- [68] International Committee of Medical Journal Editors. Available at http://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role-of-authors-and-contributors.html; accessed July 07, 2014.

#### Anney 1 PAM-13 Ougetionnaire Sample

Below are some statements that people sometimes make when they talk about their health. Please indicate how much you agree or disagree with each statement as it applies to you personally by circling your answer. Your answers should be what is true for you and not what you think others might want you to say.

If the statement does not apply to you, circle N/A.

| 1. | When all is said and done, I am the person who is responsible for taking care of my health | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
|---|---|---|---|---|---|---|
| 2. | Taking an active role in my own health care is<br>the most important thing that affects my health | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 3. | I am confident I can help prevent or reduce<br>problems associated with my health | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 4. | I know what each of my prescribed medications do | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 5. | I am confident that I can tell whether I need to<br>go to the doctor or whether I can take care of a<br>health problem myself | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 6, | I am confident that I can tell a doctor concerns I have even when he or she does not ask | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 7. | I am confident that I can follow through on<br>medical treatments I may need to do at home | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 8. | I understand my health problems and what causes them | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 9. | I know what treatments are available for my<br>health problems | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 10. | I have been able to maintain (keep up with)<br>lifestyle changes, like eating right or exercising | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 11. | I know how to prevent problems with my health | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 12. | I am confident I can figure out solutions when<br>new problems arise with my health | Disagree<br>Strongly<br>(1) | Disagree (2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |
| 13. | I am confident that I can maintain lifestyle<br>changes, like eating right and exercising, even<br>during times of stress | Disagree<br>Strongly<br>(1) | Disagree<br>(2) | Agree<br>(3) | Agree<br>Strongly<br>(4) | N/A<br>(5) |

Insignia Health. "Patient Activation Measure; Copyright<sup>©</sup> 2003-2011, University of Oregon. All Rights reserved." Contact Insignia Health at www.insigniahealth.com

DRAFT Version 0:03/CBA BG

# Annex 2. Patient Support Program (PSP) Utilization Questionnaire

| 12 weeks treatment: At Interim early post-treatment 24 weeks treatment: At Interim mid treatment vis | |
|---|---|
| Since the last visit, have you utilized any comp<br>Support Program? | oonents from the AbbVie Patient |
| □ No □ Please ignore questions below and return on nurse | questionnaire to your physician or study |
| ☐ Yes Please specify service(s) used: | |
| ☐ Personal support (e.g. Care Coach) | |
| ☐ Educational and information material (e.g. | magazines, leaflets, diaries) |
| | Usually daily<br>Several times per week<br>Usually once weekly<br>Less than once weekly |
| ☐ Additional digital and mobile resources | |
| ■ Reminders | |

## Annex 3. Patient Support Program (PSP) Utilization and Satisfaction Questionnaire

12 weeks treatment: At Interim early on-treatment visit, week 12 EoT visit and SVR 12 24 weeks treatment: At Interim early on-treatment visit, week 24 EoT visit and SVR 12 visit Since the last visit, have you utilized any components from the AbbVie Patient Support Program? □ No → Please ignore questions below and return questionnaire to your physician or study nurse ☐ Yes → What is your level of satisfaction of the AbbVie Patient Support Program in general? ☐ Very good ☐ Good □ Satisfactory ☐ Poor → Did the Program address your needs? ☐ Yes, fully ☐ Yes, mostly ☐ No Please specify service(s) used: ☐ Personal support (e.g. Care Coach) → Please specify your level of satisfaction: ☐ Very good ☐ Good □ Satisfactory ☐ Poor ☐ Educational and information material (e.g. magazines, leaflets, diaries) **X** □ Printed Please specify how often used: ☐ Usually daily ☐ Several times per week

Confidential Information

☐ Usually once weekly ☐ Less than once weekly

### Annex 4. Child-Pugh Classification of Severity of Cirrhosis

| | Points Assigned for Observed Findings | | |
|---|---|---|---|
| Parameter | 1 | 2 | 3 |
| Total bilirubin, μmol/L<br>(mg/dL) | <34.2<br>(<2) | 34.2 – 51.3<br>(2 – 3) | >51.3<br>(>3) |
| Serum albumin, g/L (g/dL) | >35<br>(>3.5) | 28 - 35<br>(2.8 - 3.5) | <28<br>(<2.8) |
| INR | <1.7 | 1.7 – 2.3 | >2.3 |
| Ascites* | None | Slight | Moderate to severe |
| Hepatic encephalopathy** | None | Grade 1 or 2<br>(or suppressed with<br>medication) | Grade 3 or 4<br>(or refractory) |

<sup>\*</sup> None.

Slight ascites = Ascites detectable only by ultrasound examination.

Moderate ascites = Ascites manifested by moderate symmetrical distension of the abdomen.

Severe ascites = Large or gross ascites with marked abdominal distension.

- \*\* Grade 0: normal consciousness, personality, neurological examination, electroencephalogram.
  - Grade 1: restless, sleep disturbed, irritable/agitated, tremor, impaired handwriting, 5 cps waves.
  - Grade 2: lethargic, time-disoriented, inappropriate behavior, asterixis, ataxia, slow triphasic waves.
  - Grade 3: somnolent, stuporous, place-disoriented, hyperactive reflexes, rigidity, slower waves.
  - Grade 4: unarousable coma, no personality/behavior, decerebrate, slow 2 to 3 cps delta activity

#### 14.0 Protocol Signature Page

# AbbVie Post Marketing Observational Study Protocol (P16-014)

Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, + Dasabuvir, ± Ribavirin and Patient Support Program in Patients with Chronic Hepatitis C - An Observational Study in Israel (CITRINE STUDY)



21 APR 2016

Date

20 Ppic 2-16

04 May 2016

may 2014